CLINICAL TRIAL: NCT03426995
Title: A Randomised, Double-blind (Sponsor Open), Placebo-controlled, Three Part Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single (in Both Fed and Fasted States) or Repeat Doses of GSK3358699 in Healthy Male Participants
Brief Title: First-time-in-Human (FTIH) Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single (in Both Fed and Fasted States) or Repeat Doses of GSK3358699
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was terminated for strategic reasons following the emergence of new data.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 207546; 2017-003997-15 (EudraCT Number)
Record Dates: First submitted 2018-02-02; First posted 2018-02-09 (Actual); Results first posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-10

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Cantharidin

STUDY DESIGN:
Intervention Model Description: Study will be conducted as Part A, B and C. Part A will consist of 2-interlocking cohorts, where each subject will receive maximum 2-single ascending oral doses of GSK3358699 and 1 dose of placebo, in Treatment Periods (TP) 1 to 3. In TP 4 subjects will receive GSK3358699, dose evaluated in TP (1 to 3) or placebo, with cantharidin induced blisters and either LPS or GM-CSF in vivo challenge. Part B will comprise of single cohort taking part in two-way cross over, with open label phase where each subject will receive single oral dose of GSK3358699 (based on Part A), under fed and fasted conditions in each TP. Part C will consist of 3 cohorts with multiple ascending doses, with every cohort having one repeat dose TP with 14 days of daily dosing of either GSK3358699 or placebo. Subjects on Day 14 will receive cantharidin induced blisters with either LPS or GM-CSF in vivo challenge. An optional, cohort 7 may be included for further dose evaluation of GSK3358699 or alternate dosing schedule.
Who Masked: Participant, Investigator
Masking Description: This will be a double blind (sponsor open) study with respect to allocation of GSK3358699 or placebo to subjects. All site staff will be blinded with the exception of un-blinded pharmacists. Investigators will be un-blinded with respect to the LPS and GM-CSF allocation. The food effect part of the study (Part B) will be open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- GSK3358699, Part A, Cohort 1 (Experimental): Part A will comprise of 4 TPs. The subjects in this cohort will receive GSK3358699, as single escalation dose, during TP (1 to 3) with planned escalated doses as 1 mg, 10 mg and 35 mg. Dose of 1 mg will be given as solution and doses of 10 mg and 35 mg, will be given as a capsule. Each TP will be of 1 day and separated by a washout Period of 14-days. Post completion of the dose-escalation TPs, an additional dosing TP 4 will be included where the subjects from each TP (1 to 3), will receive control blisters induced on forearm (0.2 % cantharidin) at Day -10. The subjects in cohort 1 will receive GSK3358699 at a dose level already given in TP 1-3, and will then receive an intravenous in vivo LPS challenge at a dose not exceeding 0.75 nanogram per kilogram post administration of GSK3358699. The subjects will then have blisters induced on the forearm approximately 20 minutes after the challenge. LPS dose will be based on data of study 207654 (NCT03306589).
  Interventions: Drug: GSK3358699; Biological: LPS; Other: Cantharidin
- GSK3358699, Part A, Cohort 2 (Experimental): Part A will comprise of 4 TPs. The subjects in this cohort will receive GSK3358699, as single escalation dose during TP (1 to 3) with planned escalated doses as 3 mg, 20 mg and 45 mg. Dose of 3 mg will be given as solution and that of 20 and 45 mg, as capsule. Each TP will be of 1 day and separated by a washout Period of 14-days. Post completion of the dose-escalation TPs, an additional dosing TP 4 will be included where the subjects from each TP (1 to 3), will receive control blisters induced on forearm (0.2 % cantharidin) at Day -10. The subjects in cohort 2 will receive GSK3358699 at a dose level already given in TP 1-3, and will then receive 60 microgram per meter^2 of in vivo GM CSF challenge as an intravenous infusion during TP 4, post administration of GSK3358699. The subjects will then have blisters induced on the forearm approximately 20 minutes after the challenge GM-CSF infusion. GM-CSF dose will be based on data of study 207654 (NCT03306589).
  Interventions: Drug: GSK3358699; Biological: GM-CSF; Other: Cantharidin
- Placebo, Part A, Cohort 1 (Placebo Comparator): Part A will comprise of 4 TPs. The subjects in this cohort will receive matching Placebo solution to the study drug GSK3358699 solution for 1 mg and a matching placebo capsule to the study drug GSK3358699, 10 mg and 35 mg capsule, during TP (1 to 3). Each TP will be of 1 day and separated by a washout Period of 14-days. Post completion of the dose-escalation TPs, an additional dosing TP 4 will be included where the subjects from each TP (1 to 3), will receive control blisters induced on forearm (0.2 % cantharidin) at Day -10. The subjects in cohort 1 will receive Placebo at a dose level already given in TP 1-3, and will then receive an intravenous in vivo LPS challenge at a dose not exceeding 0.75 nanogram per kilogram post administration of Placebo. The subjects will then have blisters induced on the forearm approximately 20 minutes after the challenge. LPS dose will be based on data of study 207654 (NCT03306589).
  Interventions: Drug: Placebo; Biological: LPS; Other: Cantharidin
- Placebo, Part A, Cohort 2 (Placebo Comparator): Part A will comprise of 4 TPs. The subjects in this cohort will receive matching Placebo solution to the study drug GSK3358699 solution for 3 mg and a matching placebo capsule to the study drug GSK3358699, for 20 and 45 mg capsule, during TP (1 to 3). Each TP will be of 1 day and separated by a washout Period of 14-days. Post completion of the dose-escalation TPs, an additional dosing TP 4 will be included where the subjects from each TP (1 to 3), will receive control blisters induced on forearm (0.2 % cantharidin) at Day -10. The subjects in cohort 2 will receive Placebo at a dose level already given in TP 1-3, and will then receive 60 microgram per meter^2 of in vivo GM CSF challenge as an intravenous infusion during TP 4, post administration of Placebo. The subjects will then have blisters induced on the forearm approximately 20 minutes after the challenge GM-CSF infusion. GM-CSF dose will be based on data of study 207654 (NCT03306589).
  Interventions: Drug: Placebo; Biological: GM-CSF; Other: Cantharidin
- Part B, GSK3358699 under Fasted followed by Fed conditions (Experimental): The subjects in this arm will receive single oral dose of GSK3358699, at a dose level evaluated in Part A, under fasted condition in TP1 followed by fed condition in TP2. This cohort intended to evaluate the effect of food.
  Interventions: Drug: GSK3358699
- Part B, GSK3358699 under Fed followed by Fasted conditions (Experimental): The subjects in this arm will receive single oral dose of GSK3358699, at a dose level evaluated in Part A, under fed condition in TP1 followed by fasted condition in TP2. This cohort intended to evaluate the effect of food.
  Interventions: Drug: GSK3358699
- GSK3358699, Part C (Experimental): The dose level for the first cohort in Part C will be decided following completion of Part A of the study for GSK3358699. The subjects in this arm will constitute 3 cohorts each (cohort 4 to 6), where the subjects will receive GSK3358699, as one repeat dose treatment once daily for 14-consecutive days. Subjects will have control blisters induced on the forearm (0.2% cantharidin) on Day -10. On the Day 14 of each cohort, each subject will receive an intravenous in vivo LPS challenge at a dose not exceeding 0.75 nanogram per kilogram or an intravenous infusion of GM-CSF, in vivo as 60 microgram per meter^2. The administration of LPS or GM CSF will be followed by blister induction on forearm (0.2 % cantharidin).
  Interventions: Drug: GSK3358699; Biological: GM-CSF; Biological: LPS; Other: Cantharidin
- Placebo, Part C (Placebo Comparator): The subjects in this cohort will receive a matching placebo to GSK3358699, Part C, as a single oral dose once daily for 14 consecutive days. The subjects in this arm will constitute 3 cohorts each (cohort 4 to 6), where the subjects will receive placebo, as one repeat dose treatment once daily for 14-consecutive days. Subjects will have control blisters induced on the forearm (0.2% cantharidin) on Day -10. On the Day 14 of each cohort, each subject will receive an intravenous in vivo LPS challenge at a dose not exceeding 0.75 nanogram per kilogram or an intravenous infusion of GM-CSF, in vivo as 60 microgram per meter^2. The administration of LPS or GM CSF will be followed by blister induction on forearm (0.2 % cantharidin).
  Interventions: Drug: Placebo; Biological: GM-CSF; Biological: LPS; Other: Cantharidin

INTERVENTIONS:
Drug: Placebo — Placebo will be administered as a matching oral solution or matching capsule to study drug GSK3358699, during Part A and C once daily
  Arms: Placebo, Part A, Cohort 1; Placebo, Part A, Cohort 2; Placebo, Part C
Drug: GSK3358699 — GSK3358699, will be administered from 1 mg to 45 mg as an oral solution (1 to 10 mg) or as a capsule (3 to 45 mg), in Part A, B and Part C once daily.
  Arms: GSK3358699, Part A, Cohort 1; GSK3358699, Part A, Cohort 2; GSK3358699, Part C; Part B, GSK3358699 under Fasted followed by Fed conditions; Part B, GSK3358699 under Fed followed by Fasted conditions
Biological: GM-CSF — The GM-CSF will be administered as an intravenous infusion to subjects as 60 microgram per meter^2 in Part A (Day 1) and Part C (Day 14).This will be administered for 2 hours approximately, no later than 24 hours post -dose of the GSK3358699 or placebo in Part C
  Arms: GSK3358699, Part A, Cohort 2; GSK3358699, Part C; Placebo, Part A, Cohort 2; Placebo, Part C
Biological: LPS — LPS will be administered as an intravenous injection to subjects not exceeding 0.75 nanogram per kilogram in Part A (Day 1) and Part C (Day 14). This will be administered no later than 24 hours post -dose of the GSK3358699 or placebo in Part C.
  Arms: GSK3358699, Part A, Cohort 1; GSK3358699, Part C; Placebo, Part A, Cohort 1; Placebo, Part C
Other: Cantharidin — This will be applied as a topical application with 0.7% cantharidin liquid which will be diluted with acetone to 0.2%.
  Arms: GSK3358699, Part A, Cohort 1; GSK3358699, Part A, Cohort 2; GSK3358699, Part C; Placebo, Part A, Cohort 1; Placebo, Part A, Cohort 2; Placebo, Part C

SUMMARY:
This FTIH study, intends to identify the doses of GSK3358699, which are well tolerated by the subjects whilst delivering a robust pharmacodynamic (PD) response. This study will evaluate the safety, tolerability, pharmacokinetic (PK) and PD profile of single (in both fed and fasted states) and multiple ascending doses of GSK3358699 in healthy male subjects within a pre-defined and controlled pharmacodynamic and pharmacokinetic range for each cohort. It also intends to understand the effect of GSK3358699 on systemic markers of inflammation following low dose in vivo lipopolysaccharide (LPS) or Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) challenge and local inflammation in cantharidin-induced blisters. The study has been carefully designed to explore the in vivo biology of the target and the potential for the study drug to become a transformative medicine for subjects in multiple immuno-inflammatory disease indications.

DETAILED DESCRIPTION:
Subjects who are enrolled in the dose escalation treatment Periods of Part A may choose to only take part in the dose escalation treatment Periods 1-3, or may choose to also take part in the challenge Treatment Period (Period 4). If a subject chooses to participate in the dose escalation treatment Periods 1-3 only, or does not (at screening) meet the eligibility criteria specific to challenges (treatment Period 4), a new subject will be recruited for treatment Period 4 only and will be regarded as a replacement subject. The study will be conducted in three Parts. Total duration for participation will be approximately 19 weeks for subjects taking part in all three dose escalation treatment Periods and 23 weeks if a subject takes part in all four treatment Periods of Part A. For replacement subjects only taking part in the challenge treatment Period (Period 4), approximate study duration will be 10 weeks. Total duration for participation will be approximately 9 weeks for Part B and 12 weeks for Part C. The study will be conducted in up to 80 subjects.

ELIGIBILITY:
Inclusion Criteria: - Subjects enrolled into the study, where they will be administered LPS or GM-CSF challenge, must be 18 to 55 years of age inclusive, at the time of signing the informed consent. Subjects enrolled into the study where they will not be administered LPS or GM-CSF challenge must be 18 to 65 years of age inclusive, at the time of signing the informed consent. - Subjects must be overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. - Body weight must be > = 50 kilogram (kg) and body mass index (BMI) within the range 18.5-35.0 kg per square meter (kg/m^2) (inclusive). - Male subjects agreeing to use contraceptive methods during the treatment Period and for at least 91 days, after the last dose of study treatment and refrain from donating sperm during this Period. - Capable of giving informed consent. Exclusion Criteria: - Current or chronic history of pancreatitis, diabetes mellitus or impaired glucose tolerance, gastrointestinal disease, liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones), anaphylaxis, and /or anaphylactoid (resembling anaphylaxis) reactions [Sampson et al 2006], cardiac disease including clinically significant ventricular arrhythmias or long QT syndrome, renal disease where clinically significant (minor abnormalities may be permitted base on discussion between investigator and medical monitor), respiratory disease or conditions including but not limited to asthma, chronic obstructive pulmonary disease (COPD), and bronchiectasis and any current respiratory infection (childhood asthma is not an exclusion criterion), sensitivity or severe allergic responses to any of the challenge agents or cantharidin, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation; frequent vasovagal syncope, surgery requiring general anaesthetic or significant trauma in 3 months leading to study enrolment, relevant skin conditions (e.g. recent history of eczema or recurrent eczema, keloid, skin allergies, psoriasis, atopic dermatitis, and vitiligo) which in the opinion of the investigator could pose safety issues or cause interference with study procedures, sepsis, coagulation disorders, peripheral edema, lymphangitis, lymphedema, pleural or pericardial effusion, hemorrhage (eg sub-arachnoid) or hemophilia or a related bleeding disorder. - History of malignancies e.g. recurrent basal cell carcinoma, hematological malignancy. - For subjects receiving cantharidin: Presence on either forearm of tattoos, naevi, hypertrophic scars, keloids, hyper- or hypo- pigmentation that may, in the opinion of the Investigator, interfere with study assessments. Subjects with very fair skin, very dark skin, excessive hair or any skin abnormalities that may, in the opinion of the Investigator, interfere with study assessments. - Family history of premature cardiovascular disease or long QT syndrome. - QT interval with Fridericia's correction (QTcF) > 450 millisecond (msec), based on averaged QTcF values of triplicate ECGs obtained over a brief recording period. - Unable or unwilling to refrain from taking prescription or non-prescription drugs (including vitamins and dietary or herbal supplements) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before the start of study treatment until completion of the follow-up visit. Paracetamol, at a dose of <= 2 grams per day was permitted for use anytime during the study. Other concomitant medications will be considered on case by case basis. - The subjects have participated in a clinical trial and received an investigational product within the following time period prior to the first dosing day in the study: 30 days; 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) or currently in a study of an investigational device. - Exposure to more than four new chemical entities within 12 months prior to the first dosing day. - Previous exposure to intravenous lipopolysaccharide (LPS) in a clinical research setting. - Alanine transaminase (ALT) >1.5x upper limit of normal (ULN) at screening. - Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) at screening. - Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. - A positive pre-study drug/alcohol screen at screening. - A positive test for human immunodeficiency virus (HIV) antibody at screening. - Persistent clinically significant abnormal C-reactive protein (CRP) levels at screening - Persistent clinically significant abnormal white cell count (WCC) levels at screening (if clinically significant abnormality is detected, WCC can be retested as clinically indicated) - Platelets < 150 x 10^9 per liter (L) at screening. - Fasted Triglycerides >3.4 millimole per liter (mmol/L) at screening. - Fasted Total cholesterol >7.7 mmol/L at screening. - Random glucose > = 11.1 mmol/L at screening. - Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening. - History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 units. One unit is equivalent to 8 gram of alcohol: a half-pint (approximately 240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL). - Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period. - Unable to comply with precautions to minimize phototoxicity risk.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available, within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided, after a research proposal is submitted and has submitted approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided, for an initial period of 12 months but an extension can be granted, when justified for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Brown JA, Bal J, Simeoni M, Williams P, Mander PK, Soden PE, Daga S, Fahy WA, Wong GK, Bloomer JC, Erwig L, Cui Y, Fernando D, Carnaghan H, Banham-Hall EJ, Hopkins S, Davis BG, Oliveira JJD, Prinjha RK. A randomized study of the safety and pharmacokinetics of GSK3358699, a mononuclear myeloid-targeted bromodomain and extra-terminal domain inhibitor. Br J Clin Pharmacol. 2022 May;88(5):2140-2155. doi: 10.1111/bcp.15137. Epub 2021 Dec 18. PMID 34773923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind, placebo-controlled, 3-part study. Part A was single ascending dose crossover with 2 interlocking cohorts(1 and 2);Part B was planned to be a single dose, open-label, 2-way crossover in fed, fasted conditions(Cohort3);Part C was repeat dose design in sequential cohorts(4,5) and cohorts 6 to 8 were planned.
Pre-assignment Details: A total 48 participants were enrolled in this study. Part B and Part C (Cohorts 6 to 8) were not initiated as the study was terminated early due to strategic reasons following emergence of new data. Hence, no participants were enrolled in Part B and Part C (Cohorts 6 to 8).
Groups:
- Part A: Cohort 1- Sequence PCEP: Participants in Part A Cohort 1 were planned to receive a single dose (SD) of placebo (Treatment P) on Day 1 in treatment Period 1. Participants were received a SD of GSK3358699 10 milligram (mg) (Treatment C) on Day 1 in treatment Period 2; followed by a SD of GSK3358699 40 mg (Treatment E) on Day 1 in treatment Period 3. On Day 1 of treatment Period 4, participants were administered a SD of placebo (Treatment P) followed by intravenous (IV) administration of in vivo lipopolysaccharide (LPS) challenge at a dose of 0.75 nanograms per kilogram (ng/kg) and further treated with 0.2 percent (%) cantharidin for induction of blisters on the forearm. GSK3358699 and placebo were administered via the oral route. There was a washout period of 14 days between each treatment period.
- Part A: Cohort 1- Sequence PCER: Participants in Part A Cohort 1 received a SD of placebo (Treatment P) on Day 1 in treatment Period 1; followed by a SD of GSK3358699 10 mg (Treatment C) on Day 1 in treatment Period 2; followed by a SD of GSK3358699 40 mg (Treatment E) on Day 1 in treatment Period 3. On Day 1 of treatment Period 4, participants were administered a SD of GSK3358699 25 mg (Treatment R) followed by IV administration of in vivo LPS challenge at a dose of 0.75 ng/kg and further treated with 0.2% cantharidin for induction of blisters on the forearm. GSK3358699 and placebo were administered via the oral route. There was a washout period of 14 days between each treatment period.
- Part A: Cohort 1- Sequence APEP: Participants in Part A Cohort 1 received a SD of GSK3358699 1 mg (Treatment A) on Day 1 in treatment Period 1; followed by a SD of placebo (Treatment P) on Day 1 in treatment Period 2; followed by a SD of GSK3358699 40 mg (Treatment E) on Day 1 in treatment Period 3. On Day 1 of treatment Period 4, participants were administered a SD of placebo (Treatment P) followed by IV administration of in vivo LPS challenge at a dose of 0.75 ng/kg and further treated with 0.2% cantharidin for induction of blisters on the forearm. GSK3358699 and placebo were administered via the oral route. There was a washout period of 14 days between each treatment period.
- Part A: Cohort 1- Sequence APER: Participants in Part A Cohort 1 received a SD of GSK3358699 1 mg (Treatment A) on Day 1 in treatment Period 1; followed by a SD of placebo (Treatment P) on Day 1 in treatment Period 2; followed by a SD of GSK3358699 40 mg (Treatment E) on Day 1 in treatment Period 3. On Day 1 of treatment Period 4, participants were administered a SD of GSK3358699 25 mg (Treatment R) followed by IV administration of in vivo LPS challenge at a dose of 0.75 ng/kg and further treated with 0.2% cantharidin for induction of blisters on the forearm. GSK3358699 and placebo were administered via the oral route. There was a washout period of 14 days between each treatment period.
- Part A: Cohort 1- Sequence ACPP: Participants in Part A Cohort 1 received a SD of GSK3358699 1 mg (Treatment A) on Day 1 in treatment Period 1; followed by a SD of GSK3358699 10 mg (Treatment C) on Day 1 in treatment Period 2; followed by a SD of placebo (Treatment P) on Day 1 in treatment Period 3. On Day 1 of treatment Period 4, participants were administered a SD of placebo (Treatment P) followed by IV administration of in vivo LPS challenge at a dose of 0.75 ng/kg and further treated with 0.2% cantharidin for induction of blisters on the forearm. GSK3358699 and placebo were administered via the oral route. There was a washout period of 14 days between each treatment period.
- Part A: Cohort 1- Sequence ACPR: Participants in Part A Cohort 1 received a SD of GSK3358699 1 mg (Treatment A) on Day 1 in treatment Period 1; followed by a SD of GSK3358699 10 mg (Treatment C) on Day 1 in treatment Period 2; followed by a SD of placebo (Treatment P) on Day 1 in treatment Period 3. On Day 1 of treatment Period 4, participants were administered a SD of GSK3358699 25 mg (Treatment R) followed by IV administration of in vivo LPS challenge at a dose of 0.75 ng/kg and further treated with 0.2% cantharidin for induction of blisters on the forearm. GSK3358699 and placebo were administered via the oral route. There was a washout period of 14 days between each treatment period.
- Part A: Cohort 2- Sequence PDFP: Participants in Part A Cohort 2 received a SD of placebo (Treatment P) on Day 1 in treatment Period 1; followed by a SD of GSK3358699 20 mg (Treatment D) on Day 1 in treatment Period 2; followed by a SD of GSK3358699 30 mg (Treatment F) on Day 1 in treatment Period 3. On Day 1 of treatment Period 4, participants were administered a SD of placebo (Treatment P) followed by IV administration of in vivo administration of Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) at a dose of 60 micrograms per meter square (mcg/m^2) and further treated with 0.2% cantharidin for induction of blisters on the forearm. GSK3358699 and placebo were administered via the oral route. There was a washout period of 14 days between each treatment period.
- Part A: Cohort 2- Sequence PDFR: Participants in Part A Cohort 2 received a SD of placebo (Treatment P) on Day 1 in treatment Period 1; followed by a SD of GSK3358699 20 mg (Treatment D) on Day 1 in treatment Period 2; followed by a SD of GSK3358699 30 mg (Treatment F) on Day 1 in treatment Period 3. On Day 1 of treatment Period 4, participants were administered a SD of GSK3358699 25 mg (Treatment R) followed by IV administration of in vivo administration of GM-CSF at a dose of 60 mcg/m^2 and further treated with 0.2% cantharidin for induction of blisters on the forearm. GSK3358699 and placebo were administered via the oral route. There was a washout period of 14 days between each treatment period.
- Part A: Cohort 2- Sequence BPFP: Participants in Part A Cohort 2 received a SD of GSK3358699 3 mg (Treatment B) on Day 1 in treatment Period 1; followed by a SD of placebo (Treatment P) on Day 1 in treatment Period 2; followed by a SD of GSK3358699 30 mg (Treatment F) on Day 1 in treatment Period 3. On Day 1 of treatment Period 4, participants were administered a SD of placebo (Treatment P) followed by IV administration of in vivo administration of GM-CSF at a dose of 60 mcg/m^2 and further treated with 0.2% cantharidin for induction of blisters on the forearm. GSK3358699 and placebo were administered via the oral route. There was a washout period of 14 days between each treatment period.
- Part A: Cohort 2- Sequence BPFR: Participants in Part A Cohort 2 were planned to receive a SD of GSK3358699 3 mg (Treatment B) on Day 1 in treatment Period 1.Participants were received a SD of placebo (Treatment P) on Day 1 in treatment Period 2; followed by a SD of GSK3358699 30 mg (Treatment F) on Day 1 in treatment Period 3. On Day 1 of treatment Period 4, participants were administered a SD of GSK3358699 25 mg (Treatment R) followed by IV administration of in vivo administration of GM-CSF at a dose of 60 mcg/m^2 and further treated with 0.2% cantharidin for induction of blisters on the forearm. GSK3358699 and placebo were administered via the oral route. There was a washout period of 14 days between each treatment period.
- Part A: Cohort 2- Sequence BDPP: Participants in Part A Cohort 2 received a SD of GSK3358699 3 mg (Treatment B) on Day 1 in treatment Period 1; followed by a SD of GSK3358699 20 mg (Treatment D) on Day 1 in treatment Period 2; followed by a SD of placebo (Treatment P) on Day 1 in treatment Period 3. On Day 1 of treatment Period 4, participants were administered a SD of placebo (Treatment P) followed by IV administration of in vivo administration of GM-CSF at a dose of 60 mcg/m^2 and further treated with 0.2% cantharidin for induction of blisters on the forearm. GSK3358699 and placebo were administered via the oral route. There was a washout period of 14 days between each treatment period.
- Part A: Cohort 2- Sequence BDPR: Participants in Part A Cohort 2 received a SD of GSK3358699 3 mg (Treatment B) on Day 1 in treatment Period 1; followed by a SD of GSK3358699 20 mg (Treatment D) on Day 1 in treatment Period 2; followed by a SD of placebo (Treatment P) on Day 1 in treatment Period 3. On Day 1 of treatment Period 4, participants were administered a SD of GSK3358699 25 mg (Treatment R) followed by IV administration of in vivo administration of GM-CSF at a dose of 60 mcg/m^2 and further treated with 0.2% cantharidin for induction of blisters on the forearm. GSK3358699 and placebo were administered via the oral route. There was a washout period of 14 days between each treatment period.
- Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted: Participants in Part B Cohort 3 were planned to receive a SD of GSK3358699 under fed conditions on Day 1 in treatment Period 1; followed by a SD of GSK3358699 under fasted conditions on Day 1 in treatment Period 2. There was a planned washout period of 14 days between each treatment period.
- Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed: Participants in Part B Cohort 3 were planned to receive a SD of GSK3358699 under fasted conditions on Day 1 in treatment Period 1; followed by a SD of GSK3358699 under fed conditions on Day 1 in treatment Period 2. There was a planned washout period of 14 days between each treatment period.
- Part C: Cohort 4 and 5- Placebo RD: Participants received once daily repeat dose (RD) of placebo on Days 1 to 14. In Cohort 4, on Day 14, participants were administered an IV in vivo LPS challenge at a dose of 0.75 ng/kg or an IV infusion of GM-CSF, in vivo at a dose of 60 mcg/m^2. The administration of LPS or GM-CSF was followed by blister induction on forearm (0.2% cantharidin).
- Part C: Cohort 4 and 5- GSK3358699 10 mg RD: Participants received once daily repeat dose of GSK3358699 10 mg on Days 1 to 14. In Cohort 4, on Day 14, participants were administered an IV in vivo LPS challenge at a dose of 0.75 ng/kg or an IV infusion of GM-CSF, in vivo at a dose of 60 mcg/m^2. The administration of LPS or GM-CSF was followed by blister induction on forearm (0.2% cantharidin).
- Part C: Cohort 6- GSK3358699 or Placebo RD: Participants in Part C Cohort 6 were planned to receive once daily repeat dose of GSK3358699 or placebo on Days 1 to 14.
- Part C: Cohort 7- GSK3358699 or Placebo RD: Participants in Part C Cohort 7 were planned to receive once daily repeat dose of GSK3358699 or placebo on Days 1 to 14.
- Part C: Cohort 8- GSK3358699 or Placebo RD: Participants in Part C Cohort 8 were planned to receive once daily repeat dose of GSK3358699 or placebo on Days 1 to 14. On Day 14, participants were planned to receive an IV in vivo LPS challenge at a dose of 0.75 ng/kg or an IV infusion of GM-CSF, in vivo as 60 mcg/m^2. The administration of LPS or GM-CSF was planned to be followed by blister induction on forearm (0.2% cantharidin).
Period: Part A: Cohort 1-Period 1 (Day1)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 0 | 2 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol defined stopping criteria | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA:Cohort1-WashoutPeriod1(Upto Day14)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 0 | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort 1-Period 2 (Day1)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 1 (New participant enrolled and dosed.) | 2 | 1 (New participant enrolled and dosed.) | 2 | 1 | 3 (Two additional participants were enrolled and dosed.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA:Cohort1-WashoutPeriod2(Upto Day14)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 1 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort 1-Period 3 (Day1)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 1 | 2 | 1 | 2 | 1 (New participant enrolled and dosed.) | 2 (New participant enrolled and dosed.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA:Cohort1-WashoutPeriod3(Upto Day14)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort 1-Period 4 (Day1)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort 2-Period 1 (Day1)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA:Cohort2-WashoutPeriod1(Upto Day14)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort 2-Period 2 (Day1)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 (Two additional participants were enrolled and dosed.) | 1 | 2 (New participant enrolled and dosed.) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA:Cohort2-WashoutPeriod2(Upto Day14)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort 2-Period 3 (Day1)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA:Cohort2-WashoutPeriod3(Upto Day14)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort 2-Period 4 (Day1)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 (New participant enrolled and dosed.) | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B: Cohort 3- Period 1 (Day 1)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartB:Cohort3-WashoutPeriod (Upto Day14)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B: Cohort 3- Period 2 (Day 1)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C: Cohorts 4 to 8 (Days 1 to 14)
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 14 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 12 | 0 | 0 | 0
Not completed — Study Closed/Terminated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 9 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated due to strategic reasons following the emergence of new data. Part B and Part C (Cohorts 6 to 8) were not initiated due to termination of the study. Hence, no participants were enrolled in Part B and Part C (Cohorts 6 to 8).
Groups:
- Part C: Cohort 4 and 5- Placebo RD: Participants received once daily RD of placebo on Days 1 to 14. In Cohort 4, on Day 14, participants were administered an IV in vivo LPS challenge at a dose of 0.75 ng/kg or an IV infusion of GM-CSF, in vivo at a dose of 60 mcg/m^2. The administration of LPS or GM-CSF was followed by blister induction on forearm (0.2% cantharidin).
- Total: Total of all reporting groups
Arm/Group | Part A: Cohort 1- Sequence PCEP | Part A: Cohort 1- Sequence PCER | Part A: Cohort 1- Sequence APEP | Part A: Cohort 1- Sequence APER | Part A: Cohort 1- Sequence ACPP | Part A: Cohort 1- Sequence ACPR | Part A: Cohort 2- Sequence PDFP | Part A: Cohort 2- Sequence PDFR | Part A: Cohort 2- Sequence BPFP | Part A: Cohort 2- Sequence BPFR | Part A: Cohort 2- Sequence BDPP | Part A: Cohort 2- Sequence BDPR | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD | Total
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 4 | 1 | 3 | 1 | 2 | 1 | 2 | 0 | 0 | 11 | 14 | 0 | 0 | 0 | 48
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  | 0 | 0 |  |  |  | 1
  >18 and <65 years | 1 | 1 | 2 | 2 | 2 | 4 | 1 | 3 | 1 | 2 | 1 | 2 |  |  | 11 | 14 |  |  |  | 47
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  | 0 | 0 |  |  |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  | 0 | 0 |  |  |  | 0
  Male | 1 | 2 | 2 | 2 | 2 | 4 | 1 | 3 | 1 | 2 | 1 | 2 |  |  | 11 | 14 |  |  |  | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 |  |  | 1 | 0 |  |  |  | 2
  White-White/Caucasian/European Heritage | 1 | 2 | 2 | 2 | 2 | 3 | 1 | 3 | 1 | 2 | 1 | 1 |  |  | 10 | 14 |  |  |  | 45
  Multiple | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 |  |  | 0 | 0 |  |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, important medical events that may jeopardize the participant or require medical or surgical intervention to prevent one of the outcomes listed before. Safety Population consisted of all randomized participants who took at least 1 dose of study treatment.
Time Frame: Up to Day 193
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Placebo SD: Participants in Part A received a SD of placebo on Day 1 in either treatment Period 1, 2 and 3. On Day 1 of treatment Period 4, participants were administered a SD of placebo followed by IV administration of in vivo LPS challenge at a dose of 0.75 ng/kg for induction of blisters on the forearm in Cohort 1 and in Cohort 2, participants were administered with IV administration of in vivo GM-CSF challenge at a dose of 60 mcg/m^2 and further treated with 0.2% cantharidin for induction of blisters on the forearm. Placebo were administered via the oral route.
- Part A: GSK3358699 1 mg SD: Participants in Part A received a SD of GSK3358699 1 mg on Day 1 in treatment Period 1.
- Part A: GSK3358699 3 mg SD: Participants in Part A received a SD of GSK3358699 3 mg on Day 1 in treatment Period 1.
- Part A: GSK3358699 10 mg SD: Participants in Part A received a SD of GSK3358699 10 mg on Day 1 in treatment Period 2.
- Part A: GSK3358699 20 mg SD: Participants in Part A received a SD of GSK3358699 20 mg on Day 1 in treatment Period 2.
- Part A: GSK3358699 25 mg SD: Participants in Part A received a SD of GSK3358699 25 mg on Day 1 in treatment Period 4. On Day 1, participants were administered a SD of GSK3358699 25 mg followed by IV administration of in vivo LPS challenge at a dose of 0.75 ng/kg for induction of blisters on the forearm in Cohort 1 and in Cohort 2, participants were administered with IV administration of in vivo GM-CSF challenge at a dose of 60 mcg/m^2 and further treated with 0.2% cantharidin for induction of blisters on the forearm. GSK3358699 were administered via the oral route.
- Part A: GSK3358699 30 mg SD: Participants in Part A received a SD of GSK3358699 30 mg on Day 1 in treatment Period 3.
- Part A: GSK3358699 40 mg SD: Participants in Part A received a SD of GSK3358699 40 mg on Day 1 in treatment Period 3.
Arm/Group | Part A: Placebo SD | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
Participants
  AEs | 8 | 2 | 3 | 2 | 3 | 8 | 4 | 3
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part B: Number of Participants With AEs and SAEs
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, important medical events that may jeopardize the participant or require medical or surgical intervention to prevent one of the outcomes listed before.
Time Frame: Up to Day 30
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Part C: Number of Participants With AEs and SAEs
Description: as for outcome 2
Time Frame: Up to Day 49
Population: Safety Population. Data was not collected for Cohorts 6 to 8 as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Number analyzed (Participants) | 11 | 14 | 0 | 0 | 0
Participants
  AEs | 7 | 8 |  |  |
  SAEs | 0 | 1 |  |  |

4. Primary Outcome: Part A: Number of Participants With Worst Case Chemistry Results by Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected for analysis of clinical chemistry parameters. PCI ranges were <30 grams per liter (g/L) (albumin), <2 or >2.75 millimoles/L (mmol/L) (calcium), >1.3* upper limit of normal (ULN) mmol/L (creatinine), <3 or >9 mmol/L (glucose), <3 or >5.5 mmol/L (potassium), and <130 or >150 mmol/L (sodium). Participants were counted in worst case category that their value changes to (low, within range or no change or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, were recorded in To within Range or No Change (NC) category. Participants were counted twice if participant had values that changed To Low and To High, so the percentages may not add to 100%.
Time Frame: Up to Day 193
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo SD | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
Participants
  Albumin: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin: To within Range or No Change | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
  Albumin: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium: To within Range or No Change | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
  Calcium: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: To within Range or No Change | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
  Creatinine: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose: To within Range or No Change | 22 | 5 | 3 | 6 | 6 | 12 | 6 | 6
  Glucose: To High | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: To within Range or No Change | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
  Potassium: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: To within Range or No Change | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
  Sodium: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Part A: Number of Participants With Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Clinical chemistry parameters assessed were alanine aminotransferase(ALT)(<10 or >50 international units per liter[IU/L]),alkaline phosphatase(ALP)(<40 or >129 IU/L),aspartate aminotransferase(AST)(<0 or >37 IU/L),cholesterol(<2.3 or >4.9 mmol/L),direct bilirubin(DB)(<0 or >5 micromoles[mcmol]/L),high density lipoprotein (DL)(<0.9 or >1.5 mmol/L),C-reactive protein(CRP)(<0.0 or >5.0mg/liter),low DL(<0 or >3.0 mmol/L), total bilirubin (<0 or >20 mcmol/L),total protein(<63 or >83 grams/L),triglycerides(<0 or >2.3 mmol/L) and blood urea nitrogen(BUN)(<4.76 or >23.24 mg/deciliter).Participants were counted in worst case category that their value changes to (low, normal or high), unless there is NC in their category.Participants whose laboratory value category was unchanged(e.g.,High to High) or whose value became normal, are recorded in "To Normal or NC" category.Participants were counted twice if participant had values that changed To Low and To High, so percentages may not add to 100%.
Time Frame: Up to Day 193
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo SD | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
Participants
  ALT: To Low,n=23,5,3,6,6,12,6,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT: To Normal or NC,n=23,5,3,6,6,12,6,6 | 22 | 5 | 3 | 6 | 6 | 12 | 6 | 6
  ALT: To High,n=23,5,3,6,6,12,6,6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALP: To Low,n=23,5,3,6,6,12,6,6 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ALP: To Normal or NC,n=23,5,3,6,6,12,6,6 | 23 | 4 | 3 | 6 | 6 | 12 | 6 | 6
  ALP: To High,n=23,5,3,6,6,12,6,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST: To Low,n=23,5,3,6,6,12,6,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST: To Normal or NC,n=23,5,3,6,6,12,6,6 | 22 | 5 | 3 | 6 | 6 | 12 | 6 | 6
  AST: To High,n=23,5,3,6,6,12,6,6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cholesterol: To Low,n=23,5,3,6,6,12,6,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cholesterol: To Normal or NC,n=23,5,3,6,6,12,6,6 | 22 | 4 | 3 | 5 | 5 | 10 | 5 | 4
  Cholesterol: To High,n=23,5,3,6,6,12,6,6 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 2
  DB: To Low,n=23,5,3,6,6,12,6,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DB:To Normal or NC,n=23,5,3,6,6,12,6,6 | 22 | 5 | 2 | 6 | 6 | 12 | 6 | 6
  DB: To High,n=23,5,3,6,6,12,6,6 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  High DL: To Low,n=23,5,3,6,6,12,6,6 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
  High DL:To Normal or NC,n=23,5,3,6,6,12,6,6 | 22 | 2 | 3 | 5 | 6 | 11 | 6 | 6
  High DL: To High,n=23,5,3,6,6,12,6,6 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  CRP: To Low,n=23,5,3,6,4,12,6,6: number analyzed (Participants) | 23 | 5 | 3 | 6 | 4 | 12 | 6 | 6
  CRP: To Low,n=23,5,3,6,4,12,6,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CRP: To Normal or NC,n=23,5,3,6,4,12,6,6: number analyzed (Participants) | 23 | 5 | 3 | 6 | 4 | 12 | 6 | 6
  CRP: To Normal or NC,n=23,5,3,6,4,12,6,6 | 18 | 5 | 2 | 6 | 4 | 4 | 6 | 5
  CRP: To High,n=23,5,3,6,4,12,6,6: number analyzed (Participants) | 23 | 5 | 3 | 6 | 4 | 12 | 6 | 6
  CRP: To High,n=23,5,3,6,4,12,6,6 | 5 | 0 | 1 | 0 | 0 | 8 | 0 | 1
  Low DL: To Low,n=23,5,3,6,6,12,6,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Low DL: To Normal or NC,n=23,5,3,6,6,12,6,6 | 21 | 5 | 2 | 4 | 5 | 11 | 5 | 4
  Low DL: To High,n=23,5,3,6,6,12,6,6 | 2 | 0 | 1 | 2 | 1 | 1 | 1 | 2
  Total bilirubin: To Low,n=23,5,3,6,6,12,6,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total bilirubin:ToNormal or NC,n=23,5,3,6,6,12,6,6 | 22 | 5 | 3 | 6 | 6 | 11 | 6 | 6
  Total bilirubin: To High,n=23,5,3,6,6,12,6,6 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Total protein: To Low,n=23,5,3,6,6,12,6,6 | 4 | 0 | 1 | 0 | 2 | 3 | 1 | 1
  Total protein:To Normal or NC,n=23,5,3,6,6,12,6,6 | 19 | 5 | 2 | 6 | 4 | 9 | 5 | 5
  Total protein: To High,n=23,5,3,6,6,12,6,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Triglycerides: To Low,n=23,5,3,6,6,12,6,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Triglycerides:To Normal or NC,n=23,5,3,6,6,12,6,6 | 17 | 3 | 2 | 4 | 4 | 12 | 3 | 4
  Triglycerides: To High,n=23,5,3,6,6,12,6,6 | 6 | 2 | 1 | 2 | 2 | 0 | 3 | 2
  BUN: To Low,n=23,5,3,6,6,12,6,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BUN: To Normal or NC,n=23,5,3,6,6,12,6,6 | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
  BUN: To High,n=23,5,3,6,6,12,6,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part B: Number of Participants With Worst Case Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline
Description: Blood samples were planned to be collected to analyze the chemistry parameters.
Time Frame: Up to Day 30
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Part B: Number of Participants With Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Blood samples were planned to be collected to analyze the chemistry parameters.
Time Frame: Up to Day 30
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Part C: Number of Participants With Worst Case Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected for analysis of chemistry parameters. PCI ranges were <30 g/L (albumin), <2 or >2.75 mmol/L (calcium), >1.3* ULN mmol/L (creatinine), <3 or >9 mmol/L (glucose), <3 or >5.5 mmol/L (potassium), and <130 or >150 mmol/L (sodium). Participants were counted in worst case category that their value changes to (low, within range or no change or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, were recorded in To within Range or No Change category. Participants were counted twice if participant had values that changed To Low and To High, so the percentages may not add to 100%.
Time Frame: Up to Day 28
Population: Safety Population. Data was not collected for Cohorts 6 to 8 as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Number analyzed (Participants) | 11 | 14 | 0 | 0 | 0
Participants
  Albumin: To Low | 0 | 0 |  |  |
  Albumin: To within Range or No Change | 11 | 14 |  |  |
  Albumin: To High | 0 | 0 |  |  |
  Calcium: To Low | 0 | 0 |  |  |
  Calcium: To within Range or No Change | 11 | 14 |  |  |
  Calcium: To High | 0 | 0 |  |  |
  Creatinine: To Low | 0 | 0 |  |  |
  Creatinine: To within Range or No Change | 11 | 14 |  |  |
  Creatinine: To High | 0 | 0 |  |  |
  Glucose: To Low | 0 | 0 |  |  |
  Glucose: To within Range or No Change | 11 | 14 |  |  |
  Glucose: To High | 0 | 0 |  |  |
  Potassium: To Low | 0 | 0 |  |  |
  Potassium: To within Range or No Change | 11 | 14 |  |  |
  Potassium: To High | 0 | 0 |  |  |
  Sodium: To Low | 0 | 0 |  |  |
  Sodium: To within Range or No Change | 11 | 14 |  |  |
  Sodium: To High | 0 | 0 |  |  |

9. Primary Outcome: Part C: Number of Participants With Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Clinical chemistry parameters assessed were ALT (<10 or >50 IU/L), ALP (<40 or >129 IU/L), AST (<0 or >37 IU/L), cholesterol (<2.3 or >4.9 mmol/L), DB (<0 or >5 mcmol/L), high DL (<0.9 or >1.5 mmol/L), CRP (<0.0 or >5.0 mg/liter), low DL (<0 or >3.0 mmol/L), total bilirubin (<0 or >20 mcmol/L), total protein (<63 or >83 grams/L), triglycerides (<0 or >2.3 mmol/L) and BUN (<4.76 or >23.24 mg/deciliter). Participants were counted in worst case category that their value changes to (low, normal or high), unless there is NC in their category. Participants whose laboratory value category was unchanged (e.g., High to High) or whose value became normal, are recorded in "To Normal or NC" category. Participants were counted twice if participant had values that changed To Low and To High, so percentages may not add to 100%.
Time Frame: Up to Day 28
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles). Data was not collected for Cohorts 6 to 8 as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Number analyzed (Participants) | 11 | 14 | 0 | 0 | 0
Participants
  ALT: To Low,n=11,14,0,0,0 | 0 | 1 |  |  |
  ALT: To Normal or NC,n=11,14,0,0,0 | 11 | 12 |  |  |
  ALT: To High,n=11,14,0,0,0 | 0 | 1 |  |  |
  ALP: To Low,n=11,14,0,0,0 | 0 | 0 |  |  |
  ALP: To Normal or NC,n=11,14,0,0,0 | 11 | 14 |  |  |
  ALP: To High,n=11,14,0,0,0 | 0 | 0 |  |  |
  AST: To Low,n=11,14,0,0,0 | 0 | 0 |  |  |
  AST: To Normal or NC,n=11,14,0,0,0 | 10 | 14 |  |  |
  AST: To High,n=11,14,0,0,0 | 1 | 0 |  |  |
  Cholesterol: To Low,n=11,14,0,0,0 | 0 | 0 |  |  |
  Cholesterol: To Normal or NC,n=11,14,0,0,0 | 9 | 13 |  |  |
  Cholesterol: To High,n=11,14,0,0,0 | 2 | 1 |  |  |
  DB: To Low,n=11,14,0,0,0 | 0 | 0 |  |  |
  DB:To Normal or NC,n=11,14,0,0,0 | 11 | 14 |  |  |
  DB: To High,n=11,14,0,0,0 | 0 | 0 |  |  |
  High DL: To Low,n=11,14,0,0,0 | 1 | 1 |  |  |
  High DL:To Normal or NC,n=11,14,0,0,0 | 10 | 13 |  |  |
  High DL: To High,n=11,14,0,0,0 | 0 | 0 |  |  |
  CRP: To Low,n=10,13,0,0,0: number analyzed (Participants) | 10 | 13 | 0 | 0 | 0
  CRP: To Low,n=10,13,0,0,0 | 0 | 0 |  |  |
  CRP: To Normal or NC,n=10,13,0,0,0: number analyzed (Participants) | 10 | 13 | 0 | 0 | 0
  CRP: To Normal or NC,n=10,13,0,0,0 | 9 | 12 |  |  |
  CRP: To High,n=10,13,0,0,0: number analyzed (Participants) | 10 | 13 | 0 | 0 | 0
  CRP: To High,n=10,13,0,0,0 | 1 | 1 |  |  |
  Low DL: To Low,n=11,14,0,0,0 | 0 | 0 |  |  |
  Low DL: To Normal or NC,n=11,14,0,0,0 | 8 | 13 |  |  |
  Low DL: To High,n=11,14,0,0,0 | 3 | 1 |  |  |
  Total bilirubin: To Low,n=11,14,0,0,0 | 0 | 0 |  |  |
  Total bilirubin:ToNormal or NC,n=11,14,0,0,0 | 11 | 14 |  |  |
  Total bilirubin: To High,n=11,14,0,0,0 | 0 | 0 |  |  |
  Total protein: To Low,n=11,14,0,0,0 | 1 | 2 |  |  |
  Total protein:To Normal or NC,n=11,14,0,0,0 | 10 | 12 |  |  |
  Total protein: To High,n=11,14,0,0,0 | 0 | 0 |  |  |
  Triglycerides: To Low,n=11,14,0,0,0 | 0 | 0 |  |  |
  Triglycerides:To Normal or NC,n=11,14,0,0,0 | 10 | 13 |  |  |
  Triglycerides: To High,n=11,14,0,0,0 | 1 | 1 |  |  |
  BUN: To Low,n=11,14,0,0,0 | 0 | 0 |  |  |
  BUN: To Normal or NC,n=11,14,0,0,0 | 11 | 14 |  |  |
  BUN: To High,n=11,14,0,0,0 | 0 | 0 |  |  |

10. Primary Outcome: Part A: Number of Participants With Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline
Description: Blood samples collected for analysis of hematology parameters. PCI ranges were >0.54 proportion of red blood cells in blood (hematocrit), >180 grams/liter (hemoglobin), <0.8 *10^9 cells/L (lymphocyte count), <1.5 *10^9 cells/L (total absolute neutrophil count [ANC]), <100 or >550 *10^9 cells/L (platelet count), and <3 or >20*10^9 cells/L (white blood cell [WBC] count). Participants were counted in worst case category that their value changes to (low, within range or no change or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, were recorded in To within Range or No Change category. Participants were counted twice if the participant had values that changed To Low and To High, so the percentages may not add to 100%.
Time Frame: Up to Day 193
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo SD | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
Participants
  Hematocrit: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit: To within Range or No Change | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
  Hematocrit: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin: To within Range or No Change | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
  Hemoglobin: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count: To Low | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Lymphocyte count: To within Range or No Change | 21 | 5 | 3 | 6 | 6 | 10 | 6 | 6
  Lymphocyte count: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet count: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet count: To within Range or No Change | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
  Platelet count: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total ANC: To Low | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Total ANC: To within Range or No Change | 23 | 4 | 3 | 6 | 6 | 12 | 6 | 6
  Total ANC: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC: To within Range or No Change | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
  WBC: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Part A: Number of Participants With Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Hematology parameters assessed were activated partial thromboplastin time (APTT) (<25 or >37 seconds), basophil count (<0.0 or >0.1*10^9 cells/L), eosinophil count (<0.0 or >0.4*10^9 cells/L), fibrinogen (<1.5 or >4.0 g/L), mean corpuscle hemoglobin (MCH) (<26.0 or >33.5 picogram), mean corpuscle volume (MCV) (<80 or >99 femtoliter), monocyte count (<0.2 or >1.0*10^9 cells/L), prothrombin time (PT) (<10 or >12 seconds), red blood cell (RBC) count (<4.4 or >5.8*10^12 cells/L) and reticulocyte count (<0.38 or >2.64 percentage of reticulocytes). Participants were counted in worst case category that their value changes to (low, normal or high), unless there is NC in their category. Participants whose laboratory value category was unchanged (e.g., High to High) or whose value became normal, are recorded in "To Normal or NC" category. Participants were counted twice if participant had values that changed To Low and To High, so percentages may not add to 100%.
Time Frame: Up to Day 193
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo SD | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
Participants
  APTT: To Low | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  APTT: To Normal or NC | 21 | 5 | 2 | 6 | 4 | 11 | 6 | 4
  APTT: To High | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Basophil count: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophil count: To Normal or NC | 23 | 5 | 3 | 6 | 5 | 12 | 6 | 6
  Basophil count: To High | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Eosinophil count: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophil count: To Normal or NC | 21 | 5 | 3 | 6 | 5 | 12 | 6 | 5
  Eosinophil count: To High | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Fibrinogen: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fibrinogen: To Normal or NC | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 5
  Fibrinogen: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  MCH: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MCH: To Normal or NC | 23 | 4 | 3 | 6 | 6 | 12 | 6 | 6
  MCH: To High | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  MCV: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MCV: To Normal or NC | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
  MCV: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Monocyte count: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Monocyte count: To Normal or NC | 19 | 5 | 3 | 6 | 6 | 6 | 6 | 6
  Monocyte count: To High | 4 | 0 | 0 | 0 | 0 | 6 | 0 | 0
  PT: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PT: To Normal or NC | 23 | 5 | 2 | 6 | 6 | 12 | 6 | 5
  PT: To High | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  RBC: To Low | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RBC: To Normal or NC | 22 | 5 | 2 | 6 | 6 | 12 | 6 | 6
  RBC: To High | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Reticulocyte count: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Reticulocyte count: To Normal or NC | 23 | 4 | 3 | 6 | 6 | 12 | 6 | 6
  Reticulocyte count: To High | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Part B: Number of Participants With Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline
Description: Blood samples were planned to be collected to analyze hematology parameters.
Time Frame: Up to Day 30
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

13. Primary Outcome: Part B: Number of Participants With Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Blood samples were planned to be collected to analyze hematology parameters.
Time Frame: Up to Day 30
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

14. Primary Outcome: Part C: Number of Participants With Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected for analysis of hematology parameters. PCI ranges were >0.54 proportion of red blood cells in blood (hematocrit), >180 grams/liter (hemoglobin), <0.8*10^9 cells/L (lymphocyte count), <1.5*10^9 cells/L (total ANC), <100 or >550*10^9 cells/L (platelet count), and <3 or >20*10^9 cells/L (WBC count). Participants were counted in worst case category that their value changes to (low, within range or no change or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, were recorded in To within Range or No Change category. Participants were counted twice if the participant had values that changed To Low and To High, so the percentages may not add to 100%.
Time Frame: Up to Day 28
Population: Safety Population. Data was not collected for Cohorts 6 to 8 as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Number analyzed (Participants) | 11 | 14 | 0 | 0 | 0
Participants
  Hematocrit: To Low | 0 | 0 |  |  |
  Hematocrit: To within Range or No Change | 11 | 14 |  |  |
  Hematocrit: To High | 0 | 0 |  |  |
  Hemoglobin: To Low | 0 | 0 |  |  |
  Hemoglobin: To within Range or No Change | 11 | 14 |  |  |
  Hemoglobin: To High | 0 | 0 |  |  |
  Lymphocyte count: To Low | 1 | 0 |  |  |
  Lymphocyte count: To within Range or No Change | 10 | 14 |  |  |
  Lymphocyte count: To High | 0 | 0 |  |  |
  Platelet count: To Low | 0 | 0 |  |  |
  Platelet count: To within Range or No Change | 11 | 14 |  |  |
  Platelet count: To High | 0 | 0 |  |  |
  Total ANC: To Low | 1 | 0 |  |  |
  Total ANC: To within Range or No Change | 10 | 14 |  |  |
  Total ANC: To High | 0 | 0 |  |  |
  WBC: To Low | 1 | 1 |  |  |
  WBC: To within Range or No Change | 10 | 13 |  |  |
  WBC: To High | 0 | 0 |  |  |

15. Primary Outcome: Part C: Number of Participants With Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Hematology parameters assessed were APTT (<25 or >37 seconds), basophil count (<0.0 or >0.1*10^9 cells/L), eosinophil count (<0.0 or >0.4*10^9 cells/L), fibrinogen (<1.5 or >4.0 g/L), MCH (<26.0 or >33.5 picogram), MCV (<80 or >99 femtoliter), monocyte count (<0.2 or >1.0*10^9 cells/L), PT (<10 or >12 seconds), RBC count (<4.4 or >5.8*10^12 cells/L) and reticulocyte count (<0.38 or >2.64 percentage of reticulocytes). Participants were counted in worst case category that their value changes to (low, normal or high), unless there is NC in their category. Participants whose laboratory value category was unchanged (e.g., High to High) or whose value became normal, are recorded in "To Normal or NC" category. Participants were counted twice if participant had values that changed To Low and To High, so percentages may not add to 100%.
Time Frame: Up to Day 28
Population: Safety Population. Data was not collected for Cohorts 6 to 8 as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Number analyzed (Participants) | 11 | 14 | 0 | 0 | 0
Participants
  APTT: To Low | 1 | 0 |  |  |
  APTT: To Normal or NC | 10 | 13 |  |  |
  APTT: To High | 0 | 1 |  |  |
  Basophil count: To Low | 0 | 0 |  |  |
  Basophil count: To Normal or NC | 11 | 14 |  |  |
  Basophil count: To High | 0 | 0 |  |  |
  Eosinophil count: To Low | 0 | 0 |  |  |
  Eosinophil count: To Normal or NC | 11 | 14 |  |  |
  Eosinophil count: To High | 0 | 0 |  |  |
  Fibrinogen: To Low | 0 | 0 |  |  |
  Fibrinogen: To Normal or NC | 11 | 14 |  |  |
  Fibrinogen: To High | 0 | 0 |  |  |
  MCH: To Low | 0 | 0 |  |  |
  MCH: To Normal or NC | 11 | 14 |  |  |
  MCH: To High | 0 | 0 |  |  |
  MCV: To Low | 0 | 0 |  |  |
  MCV: To Normal or NC | 11 | 14 |  |  |
  MCV: To High | 0 | 0 |  |  |
  Monocyte count: To Low | 0 | 0 |  |  |
  Monocyte count: To Normal or NC | 11 | 14 |  |  |
  Monocyte count: To High | 0 | 0 |  |  |
  PT: To Low | 0 | 0 |  |  |
  PT: To Normal or NC | 10 | 14 |  |  |
  PT: To High | 1 | 0 |  |  |
  RBC: To Low | 0 | 1 |  |  |
  RBC: To Normal or NC | 11 | 13 |  |  |
  RBC: To High | 0 | 0 |  |  |
  Reticulocyte count: To Low | 0 | 0 |  |  |
  Reticulocyte count: To Normal or NC | 11 | 14 |  |  |
  Reticulocyte count: To High | 0 | 0 |  |  |

16. Primary Outcome: Part A: Number of Participants With Abnormal Urinalysis Parameters
Description: Urine samples were collected from participants for analyzing the following urine parameters: potential of hydrogen (pH) and glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocytes levels by dipstick. Urine samples showing any abnormality were sent for microscopic examination to detect the presence of RBC, WBC, cellular casts, granular casts, hyaline casts, and were counted as cells per high-power field (cells/HPF). Number of participants with abnormal urinalysis result by microscopic examination have been presented.
Time Frame: Up to Day 193
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo SD | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
Participants
  RBC | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  WBC | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cellular casts | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Granular casts | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyaline casts | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Primary Outcome: Part B: Number of Participants With Abnormal Urinalysis Parameters
Description: Urine samples were planned to be collected to analyze urine parameters.
Time Frame: Up to Day 30
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

18. Primary Outcome: Part C: Number of Participants With Abnormal Urinalysis Parameters
Description: Urine samples were collected from participants for analyzing the following urine parameters: pH and glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocytes levels by dipstick. Urine samples showing any abnormality were sent for microscopic examination to detect the presence of RBC, WBC, cellular casts, granular casts, hyaline casts, and were counted as cells/HPF. Number of participants with abnormal urinalysis result by microscopic examination have been presented.
Time Frame: Up to Day 28
Population: Safety Population. Data was not collected for Cohorts 6 to 8 as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Number analyzed (Participants) | 11 | 14 | 0 | 0 | 0
Participants
  RBC | 0 | 0 |  |  |
  WBC | 1 | 1 |  |  |
  Cellular casts | 0 | 0 |  |  |
  Granular casts | 0 | 0 |  |  |
  Hyaline casts | 0 | 0 |  |  |

19. Primary Outcome: Part A: Number of Participants With Worst Case Vital Sign Results by PCI Criteria Post-Baseline Relative to Baseline
Description: Vital signs included systolic blood pressure(SBP), diastolic blood pressure(DBP), heart rate, respiratory rate and body temperature and were measured in a semi-supine position after 5 minutes rest. PCI ranges were, SBP (millimeters of mercury [mmHg]): <85 (low) or >160 (high), DBP (mmHg): <45 (low) or >100 (high), heart rate (beats per minute): <40 (low) or >110 (high), respiration rate (breaths per minute): <11(low) or >20(high) and body temperature (degrees Celsius) <35.5 (low) or >38.0 (high). Participants were counted in the worst case category that their value changes to (low, within range or no change, or high), unless there is no change in their category. Participants whose vital signs value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the "To within Range or No Change" category. Participants were counted twice if the participant had values that changed "To Low" and "To High", so the percentages may not add to 100%.
Time Frame: Up to Day 193
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo SD | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
Participants
  SBP: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP: To within Range or No Change | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
  SBP: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP: To within Range or No Change | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
  DBP: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Heart rate: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Heart rate: To within Range or No Change | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
  Heart rate: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory rate: To Low | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Respiratory rate: To within Range or No Change | 22 | 5 | 3 | 6 | 6 | 11 | 6 | 6
  Respiratory rate: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Body temperature: To Low | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Body temperature: To within Range or No Change | 22 | 5 | 3 | 5 | 6 | 11 | 6 | 6
  Body temperature: To High | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

20. Primary Outcome: Part B: Number of Participants With Worst Case Vital Sign Results by PCI Criteria Post-Baseline Relative to Baseline
Description: Vital signs were planned to be measured in a semi-supine position after 5 minutes of rest.
Time Frame: Up to Day 30
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

21. Primary Outcome: Part C: Number of Participants With Worst Case Vital Sign Results by PCI Criteria Post-Baseline Relative to Baseline
Description: Vital signs included SBP, DBP, heart rate, respiratory rate and body temperature and were measured in a semi-supine position after 5 minutes rest. PCI ranges were, SBP (mmHg): <85 (low) or >160 (high), DBP (mmHg): <45 (low) or >100 (high), heart rate (beats per minute): <40 (low) or >110 (high), respiration rate (breaths per minute): <11 (low) or >20 (high) and body temperature (degrees Celsius) <35.5 (low) or >38.0 (high). Participants were counted in the worst case category that their value changes to (low, within range or no change, or high), unless there is no change in their category. Participants whose vital signs value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the "To within Range or No Change" category. Participants were counted twice if the participant had values that changed "To Low" and "To High", so the percentages may not add to 100%.
Time Frame: Up to Day 49
Population: Safety Population. Data was not collected for Cohorts 6 to 8 as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Number analyzed (Participants) | 11 | 14 | 0 | 0 | 0
Participants
  SBP: To Low | 0 | 0 |  |  |
  SBP: To within Range or No Change | 11 | 14 |  |  |
  SBP: To High | 0 | 0 |  |  |
  DBP: To Low | 0 | 0 |  |  |
  DBP: To within Range or No Change | 11 | 14 |  |  |
  DBP: To High | 0 | 0 |  |  |
  Heart rate: To Low | 0 | 1 |  |  |
  Heart rate: To within Range or No Change | 10 | 13 |  |  |
  Heart rate: To High | 1 | 0 |  |  |
  Respiratory rate: To Low | 1 | 1 |  |  |
  Respiratory rate: To within Range or No Change | 9 | 13 |  |  |
  Respiratory rate: To High | 1 | 0 |  |  |
  Body temperature: To Low | 0 | 0 |  |  |
  Body temperature: To within Range or No Change | 11 | 14 |  |  |
  Body temperature: To High | 0 | 0 |  |  |

22. Primary Outcome: Part A: Number of Participants With Worst Case Post-Baseline Abnormal Electrocardiogram (ECG) Findings
Description: Twelve lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and QT interval corrected using the Fridericia's formula (QTcF) intervals. Abnormal findings were categorized as clinically significant (CS) and not clinically significant (NCS). Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for number of participants with worst case post-Baseline abnormal ECG findings have been presented.
Time Frame: Up to Day 193
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo SD | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 23 | 5 | 3 | 6 | 6 | 12 | 6 | 6
Participants
  Abnormal - not clinically significant | 6 | 1 | 0 | 0 | 3 | 2 | 3 | 0
  Abnormal - clinically significant | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Primary Outcome: Part B: Number of Participants With Worst Case Post-Baseline Abnormal ECG Findings
Description: Twelve lead ECGs were planned to be performed to measure PR interval, QRS duration, QT interval and QTcF.
Time Frame: Up to Day 30
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

24. Primary Outcome: Part C: Number of Participants With Worst Case Post-Baseline Abnormal ECG Findings
Description: Twelve lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and QTcF intervals. Abnormal findings were categorized as clinically significant and not clinically significant. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for number of participants with worst case post-Baseline abnormal ECG findings have been presented.
Time Frame: Up to Day 28
Population: Safety Population. Data was not collected for Cohorts 6 to 8 as no participants were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Number analyzed (Participants) | 11 | 14 | 0 | 0 | 0
Participants
  Abnormal - not clinically significant | 2 | 3 |  |  |
  Abnormal - clinically significant | 0 | 1 |  |  |

25. Secondary Outcome: Part A: Plasma Concentrations of GSK3358699
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3358699. Pharmacokinetic (PK) parameters were calculated using standard non-compartmental analysis. PK Population consisted of all participants in the Safety Population who received an active dose and for whom a PK sample was obtained and analyzed.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Median (Full Range); unit: Nanogram per milliliter
Arm/Group | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 5 | 3 | 6 | 6 | 12 | 6 | 6
Nanogram per milliliter
  Pre-dose, n=5,3,6,6,12,6,6 | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.0000 to 0.000] | 0.0000 [0.0000 to 0.0000] | 0.0000 [0.0000 to 0.0000] | 0.0000 [0.0000 to 0.0000]
  15 minutes, n=5,3,6,6,12,6,6 | 0.4950 [0.000 to 1.921] | 0.6470 [0.431 to 1.142] | 1.0480 [0.000 to 10.565] | 0.5390 [0.000 to 16.637] | 0.2620 [0.000 to 15.086] | 5.8460 [0.189 to 21.540] | 0.9245 [0.000 to 3.315]
  30 minutes, n=5,3,6,6,12,6,6 | 0.6840 [0.497 to 1.106] | 1.9510 [1.094 to 2.411] | 6.4560 [3.010 to 10.780] | 5.1050 [1.017 to 28.795] | 5.9130 [0.726 to 22.813] | 64.4810 [8.884 to 99.800] | 33.2120 [1.966 to 211.754]
  1 hour, n=5,3,6,6,12,6,6 | 0.4210 [0.264 to 0.553] | 0.9960 [0.893 to 1.440] | 3.5150 [1.234 to 8.072] | 9.1840 [4.283 to 18.108] | 11.0785 [2.165 to 17.950] | 28.4500 [20.421 to 92.656] | 28.8380 [15.838 to 39.777]
  2 hours, n=5,3,6,6,12,6,6 | 0.1810 [0.119 to 0.215] | 0.4790 [0.284 to 0.651] | 1.6930 [0.638 to 2.067] | 4.8100 [2.093 to 8.048] | 6.9495 [3.397 to 26.662] | 10.6550 [6.792 to 18.163] | 8.6735 [7.895 to 18.906]
  4 hours, n=5,2,6,6,12,6,6: number analyzed (Participants) | 5 | 2 | 6 | 6 | 12 | 6 | 6
  4 hours, n=5,2,6,6,12,6,6 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | 0.1560 [0.151 to 0.161] | 0.5265 [0.358 to 0.916] | 1.2865 [0.746 to 1.599] | 1.9095 [1.158 to 4.344] | 3.6390 [1.706 to 4.101] | 2.5920 [1.886 to 4.266]
  6 hours, n=5,3,6,6,12,6,6 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | 0.3160 [0.243 to 0.792] | 0.6720 [0.385 to 1.327] | 1.1020 [0.409 to 2.342] | 1.4305 [0.916 to 3.954] | 1.2515 [0.980 to 1.748]
  8 hours, n=5,3,6,6,12,6,6 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | 0.2120 [0.110 to 0.426] | 0.3775 [0.209 to 0.611] | 0.5915 [0.230 to 1.131] | 0.8340 [0.318 to 1.720] | 0.6665 [0.434 to 1.033]
  12 hours, n=5,3,2,6,12,6,6: number analyzed (Participants) | 5 | 3 | 2 | 6 | 12 | 6 | 6
  12 hours, n=5,3,2,6,12,6,6 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | 0.1390 [0.136 to 0.142] | 0.1490 [0.100 to 0.159] | 0.2510 [0.145 to 0.605] | 0.5195 [0.291 to 0.745] | 0.4255 [0.145 to 0.939]
  24 hours, n=5,3,6,6,9,4,5: number analyzed (Participants) | 5 | 3 | 6 | 6 | 9 | 4 | 5
  24 hours, n=5,3,6,6,9,4,5 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | 0.1510 [0.000 to 0.369] | 0.1250 [0.000 to 0.485] | 0.2090 [0.000 to 0.287]
  48 hours, n=5,3,6,6,6,6,6: number analyzed (Participants) | 5 | 3 | 6 | 6 | 6 | 6 | 6
  48 hours, n=5,3,6,6,6,6,6 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | 0.0000 [0.000 to 0.114] | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification.

26. Secondary Outcome: Part B: Plasma Concentrations of GSK3358699
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3358699.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Part C: Plasma Concentrations of GSK3358699
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3358699. PK parameters were calculated using standard non-compartmental analysis.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12 and 24 hours; Days 4, 8 and 12: Pre-dose; Day 14: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose
Population: PK Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles). Data was not collected for Cohorts 6 to 8 as no participants were enrolled.
Measure: Median (Full Range); unit: Nanogram per milliliter
Groups:
- Part C: Cohort 6- GSK3358699 RD: Participants in Part C Cohort 6 were planned to receive once daily repeat dose of GSK3358699 on Days 1 to 14.
- Part C: Cohort 7- GSK3358699 RD: Participants in Part C Cohort 7 were planned to receive once daily repeat dose of GSK3358699 on Days 1 to 14.
- Part C: Cohort 8- GSK3358699 RD: Participants in Part C Cohort 8 were planned to receive once daily repeat dose of GSK3358699 on Days 1 to 14. On Day 14, participants were planned to receive an IV in vivo LPS challenge at a dose of 0.75 ng/kg or an IV infusion of GM-CSF, in vivo as 60 mcg/m^2. The administration of LPS or GM-CSF was planned to be followed by blister induction on forearm (0.2% cantharidin).
Arm/Group | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 RD | Part C: Cohort 7- GSK3358699 RD | Part C: Cohort 8- GSK3358699 RD
Number analyzed (Participants) | 14 | 0 | 0 | 0
Nanogram per milliliter
  Day 1:Pre-dose,n=14,0,0,0 | 0.0000 [0.000 to 0.000] |  |  |
  Day 1:15 minutes,n=14,0,0,0 | 0.2825 [0.000 to 13.601] |  |  |
  Day 1:30 minutes,n=14,0,0,0 | 5.7430 [0.914 to 16.960] |  |  |
  Day 1:1 hour,n=14,0,0,0 | 3.8955 [1.758 to 12.384] |  |  |
  Day 1:2 hours,n=14,0,0,0 | 1.3365 [0.826 to 4.710] |  |  |
  Day 1:4 hours,n=14,0,0,0 | 0.5730 [0.205 to 0.922] |  |  |
  Day 1:6 hours,n=14,0,0,0 | 0.2940 [0.109 to 0.500] |  |  |
  Day 1:8 hours,n=10,0,0,0: number analyzed (Participants) | 10 | 0 | 0 | 0
  Day 1:8 hours,n=10,0,0,0 | 0.1690 [0.109 to 0.384] |  |  |
  Day 1:12 hours,n=3,0,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0
  Day 1:12 hours,n=3,0,0,0 | 0.1390 [0.120 to 0.144] |  |  |
  Day 1:24 hours,n=14,0,0,0 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. |  |  |
  Day 4: Pre-dose,n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 4: Pre-dose,n=1,0,0,0 | 0.0000 [0.000 to 0.000] |  |  |
  Day 8: Pre-dose,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 8: Pre-dose,n=2,0,0,0 | 0.0000 [0.000 to 0.000] |  |  |
  Day 12: Pre-dose,n=4,0,0,0: number analyzed (Participants) | 4 | 0 | 0 | 0
  Day 12: Pre-dose,n=4,0,0,0 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. |  |  |
  Day 14:Pre-dose,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:Pre-dose,n=2,0,0,0 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. |  |  |
  Day 14:15 minutes,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:15 minutes,n=2,0,0,0 | 4.3390 [1.836 to 6.842] |  |  |
  Day 14:30 minutes,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:30 minutes,n=2,0,0,0 | 6.0065 [4.658 to 7.355] |  |  |
  Day 14:1 hour,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:1 hour,n=2,0,0,0 | 3.0170 [2.233 to 3.801] |  |  |
  Day 14:2 hours,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:2 hours,n=2,0,0,0 | 1.4905 [0.979 to 2.002] |  |  |
  Day 14:4 hours,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:4 hours,n=2,0,0,0 | 0.8295 [0.754 to 0.905] |  |  |
  Day 14:6 hours,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:6 hours,n=2,0,0,0 | 0.6360 [0.313 to 0.959] |  |  |
  Day 14:8 hours,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:8 hours,n=2,0,0,0 | 0.3920 [0.155 to 0.629] |  |  |
  Day 14:12 hours,n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 14:12 hours,n=1,0,0,0 | 0.2730 [0.273 to 0.273] |  |  |
  Day 14:24 hours,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:24 hours,n=2,0,0,0 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. |  |  |
  Day 14:48 hours,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:48 hours,n=2,0,0,0 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. |  |  |

28. Secondary Outcome: Part A: Area Under the Plasma Concentration Curve From Time Zero to Last Time of Quantifiable Concentration (AUC[0-t]) of GSK3358699
Description: as for outcome 27
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population.
Measure: Median (Full Range); unit: Hours*nanogram per milliliter
Arm/Group | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 5 | 3 | 6 | 6 | 12 | 6 | 6
Hours*nanogram per milliliter | 0.74 [0.6 to 1.3] | 2.33 [1.7 to 2.8] | 10.77 [5.1 to 16.4] | 23.40 [18.1 to 30.5] | 31.88 [27.2 to 56.0] | 66.38 [54.6 to 128.1] | 58.09 [48.1 to 114.3]

29. Secondary Outcome: Part B: AUC(0-t) of GSK3358699
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3358699.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Part C: AUC(0-t) of GSK3358699
Description: as for outcome 27
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12 and 24 hours; Day 14: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose
Population: as for outcome 27
Measure: Median (Full Range); unit: Hours*nanogram per milliliter
Arm/Group | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 RD | Part C: Cohort 7- GSK3358699 RD | Part C: Cohort 8- GSK3358699 RD
Number analyzed (Participants) | 14 | 0 | 0 | 0
Hours*nanogram per milliliter
  Day 1, n=14,0,0,0 | 9.47 [4.8 to 20.9] |  |  |
  Day 14, n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14, n=2,0,0,0 | 11.70 [7.6 to 15.8] |  |  |

31. Secondary Outcome: Part A: Area Under the Plasma Concentration Curve From Time Zero to Infinity (AUC[0-infinity]) of GSK3358699
Description: as for outcome 27
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours*nanogram per milliliter
Arm/Group | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 5 | 3 | 5 | 6 | 9 | 4 | 5
Hours*nanogram per milliliter | NA [NA to NA] — AUC(0-infinity) could not be calculated as we need at least 3 data points in terminal elimination phase within same participant and this criteria could not be fulfilled due to insufficient data above limit of quantification (in all participants). | NA [NA to NA] — AUC(0-infinity) could not be calculated as we need at least 3 data points in terminal elimination phase within same participant and this criteria could not be fulfilled due to insufficient data above limit of quantification (in all participants). | 13.20 [5.6 to 17.0] | 23.89 [18.6 to 31.0] | 33.22 [28.4 to 57.0] | 69.13 [56.6 to 129.0] | 59.68 [49.2 to 114.7]

32. Secondary Outcome: Part B: AUC(0-infinity) of GSK3358699
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3358699.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Part C: AUC(0-infinity) of GSK3358699
Description: as for outcome 27
Time Frame: as for outcome 30
Population: as for outcome 27
Measure: Median (Full Range); unit: Hours*nanogram per milliliter
Arm/Group | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 RD | Part C: Cohort 7- GSK3358699 RD | Part C: Cohort 8- GSK3358699 RD
Number analyzed (Participants) | 7 | 0 | 0 | 0
Hours*nanogram per milliliter
  Day 1, n=7,0,0,0 | 9.07 [5.9 to 16.9] |  |  |
  Day 14, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0

34. Secondary Outcome: Part A: Area Under the Plasma Concentration Curve From Time Zero to 24 Hours (AUC[0-24]) of GSK3358699
Description: as for outcome 27
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours*nanogram per milliliter
Arm/Group | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 5 | 3 | 5 | 6 | 10 | 5 | 6
Hours*nanogram per milliliter | NA [NA to NA] — AUC(0-24) could not be calculated as we need at least 3 data points in terminal elimination phase within same participant and this criteria could not be fulfilled due to insufficient data above limit of quantification (in all participants). | NA [NA to NA] — AUC(0-24) could not be calculated as we need at least 3 data points in terminal elimination phase within same participant and this criteria could not be fulfilled due to insufficient data above limit of quantification (in all participants). | 13.17 [5.6 to 16.9] | 23.86 [18.6 to 31.0] | 32.69 [25.4 to 56.0] | 67.38 [56.4 to 128.1] | 59.05 [48.1 to 114.7]

35. Secondary Outcome: Part B: AUC(0-24) of GSK3358699
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3358699.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Part C: AUC(0-24) of GSK3358699
Description: as for outcome 27
Time Frame: Days 1 and 14: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, and 24 hours post-dose
Population: as for outcome 27
Measure: Median (Full Range); unit: Hours*nanogram per milliliter
Arm/Group | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 RD | Part C: Cohort 7- GSK3358699 RD | Part C: Cohort 8- GSK3358699 RD
Number analyzed (Participants) | 7 | 0 | 0 | 0
Hours*nanogram per milliliter
  Day 1, n=7,0,0,0 | 9.07 [5.8 to 16.9] |  |  |
  Day 14, n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 14, n=1,0,0,0 | 7.99 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual AUC(0-24) for this single participant. |  |  |

37. Secondary Outcome: Part A: Maximum Plasma Concentration (Cmax) of GSK3358699
Description: as for outcome 27
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population.
Measure: Median (Full Range); unit: Nanogram per milliliter
Arm/Group | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 5 | 3 | 6 | 6 | 12 | 6 | 6
Nanogram per milliliter | 0.68 [0.5 to 1.9] | 1.95 [1.4 to 2.4] | 6.46 [3.0 to 10.8] | 16.10 [9.1 to 28.8] | 17.47 [7.5 to 26.7] | 64.48 [20.4 to 99.8] | 34.58 [20.4 to 211.8]

38. Secondary Outcome: Part B: Cmax of GSK3358699
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3358699.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: Part C: Cmax of GSK3358699
Description: as for outcome 27
Time Frame: as for outcome 30
Population: as for outcome 27
Measure: Median (Full Range); unit: Nanogram per milliliter
Groups:
- Part C: Cohort 8- GSK3358699 RD: Participants in Part C Cohort 8 were planned to receive once daily repeat dose of GSK3358699 on Days 1 to 14. On Day 14, participants were planned to receive an IV in vivo LPS challenge at a dose of 0.75 ng/kg or an IV infusion of GM-CSF, in vivo as 60 mcg/m^2. The administration of LPS or GM CSF was planned to be followed by blister induction on forearm (0.2% cantharidin).
Arm/Group | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 RD | Part C: Cohort 7- GSK3358699 RD | Part C: Cohort 8- GSK3358699 RD
Number analyzed (Participants) | 14 | 0 | 0 | 0
Nanogram per milliliter
  Day 1, n=14,0,0,0 | 6.19 [2.6 to 17.0] |  |  |
  Day 14, n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14, n=2,0,0,0 | 6.01 [4.7 to 7.4] |  |  |

40. Secondary Outcome: Part A: Time to Cmax (Tmax) of GSK3358699
Description: as for outcome 27
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 5 | 3 | 6 | 6 | 12 | 6 | 6
Hours | 0.50 [0.3 to 1.0] | 0.50 [0.5 to 1.0] | 0.50 [0.5 to 0.5] | 1.00 [0.3 to 1.0] | 1.00 [0.2 to 2.0] | 0.76 [0.5 to 1.0] | 0.51 [0.5 to 1.1]

41. Secondary Outcome: Part B: Tmax of GSK3358699
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3358699.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

42. Secondary Outcome: Part C: Tmax of GSK3358699
Description: as for outcome 27
Time Frame: as for outcome 30
Population: as for outcome 27
Measure: Median (Full Range); unit: Hours
Arm/Group | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 RD | Part C: Cohort 7- GSK3358699 RD | Part C: Cohort 8- GSK3358699 RD
Number analyzed (Participants) | 14 | 0 | 0 | 0
Hours
  Day 1, n=14,0,0,0 | 0.50 [0.3 to 2.0] |  |  |
  Day 14, n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14, n=2,0,0,0 | 0.53 [0.5 to 0.6] |  |  |

43. Secondary Outcome: Part A: Apparent Terminal Phase Half-life (t1/2) of GSK3358699
Description: as for outcome 27
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 5 | 3 | 5 | 6 | 9 | 4 | 5
Hours | NA [NA to NA] — t1/2 could not be calculated as we need at least 3 time points in terminal elimination phase within the same participant and this criteria could not be fulfilled due to insufficient data above limit of quantification (in all participants). | NA [NA to NA] — t1/2 could not be calculated as we need at least 3 time points in terminal elimination phase within the same participant and this criteria could not be fulfilled due to insufficient data above limit of quantification (in all participants). | 2.44 [2.0 to 2.8] | 2.75 [2.0 to 3.4] | 6.02 [2.1 to 18.4] | 4.77 [3.5 to 11.8] | 6.88 [2.1 to 11.1]

44. Secondary Outcome: Part B: t1/2 of GSK3358699
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3358699.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

45. Secondary Outcome: Part C: t1/2 of GSK3358699
Description: as for outcome 27
Time Frame: as for outcome 30
Population: as for outcome 27
Measure: Median (Full Range); unit: Hours
Arm/Group | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 RD | Part C: Cohort 7- GSK3358699 RD | Part C: Cohort 8- GSK3358699 RD
Number analyzed (Participants) | 7 | 0 | 0 | 0
Hours
  Day 1, n=7,0,0,0 | 2.47 [1.4 to 3.0] |  |  |
  Day 14, n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 14, n=1,0,0,0 | 1.57 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual t1/2 for this single participant. |  |  |

46. Secondary Outcome: Part A: Plasma Concentrations of GSK3206944
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3206944. PK parameters were calculated using standard non-compartmental analysis. GSK3206944 is a metabolite of GSK3358699.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population.
Measure: Median (Full Range); unit: Nanogram per milliliter
Arm/Group | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 5 | 3 | 6 | 6 | 12 | 6 | 6
Nanogram per milliliter
  Pre-dose | 0.0000 [0.000 to 0.000] | 0.000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000] | 0.0000 [0.000 to 0.000]
  15 minutes | 0.2050 [0.000 to 0.870] | 0.2070 [0.107 to 0.247] | 0.0550 [0.000 to 0.973] | 0.0000 [0.000 to 0.292] | 0.0000 [0.000 to 6.579] | 0.0575 [0.000 to 1.462] | 0.0000 [0.000 to 0.155]
  30 minutes | 1.2090 [0.223 to 3.045] | 1.8410 [0.705 to 2.156] | 3.1930 [2.030 to 9.850] | 1.8370 [0.000 to 10.528] | 4.3810 [0.216 to 25.498] | 17.2245 [1.546 to 27.299] | 6.3350 [0.412 to 46.595]
  1 hour | 3.0310 [1.808 to 4.898] | 4.2200 [2.505 to 6.026] | 17.1455 [6.453 to 26.263] | 26.1280 [18.350 to 43.603] | 33.6145 [2.943 to 68.271] | 89.1965 [16.207 to 205.963] | 74.5130 [26.229 to 205.962]
  2 hours | 3.2830 [2.145 to 4.324] | 5.5640 [4.837 to 7.256] | 17.6535 [7.569 to 30.510] | 46.4250 [27.542 to 82.343] | 70.4010 [20.386 to 105.133] | 102.0865 [51.492 to 161.313] | 121.2220 [88.345 to 231.739]
  4 hours | 1.9110 [1.223 to 2.658] | 3.2490 [2.951 to 3.733] | 10.6790 [7.400 to 15.516] | 22.6925 [13.453 to 50.059] | 46.8165 [28.244 to 78.533] | 51.7230 [40.674 to 84.834] | 69.2315 [46.996 to 132.904]
  6 hours | 0.9490 [0.529 to 1.342] | 1.5760 [1.532 to 1.877] | 6.7745 [4.726 to 9.175] | 13.7955 [10.716 to 28.908] | 23.1275 [15.320 to 44.082] | 30.4690 [23.891 to 34.815] | 36.8305 [19.883 to 59.881]
  8 hours | 0.5840 [0.303 to 0.945] | 1.0200 [1.019 to 1.096] | 4.6515 [2.297 to 5.599] | 8.3535 [6.187 to 14.398] | 13.7165 [9.459 to 21.878] | 16.5795 [10.812 to 21.258] | 18.4825 [12.948 to 31.766]
  12 hours | 0.2540 [0.122 to 0.353] | 0.4670 [0.336 to 0.667] | 1.8400 [0.785 to 2.418] | 3.4535 [2.385 to 4.611] | 5.3830 [3.258 to 9.084] | 6.7365 [4.811 to 8.739] | 8.7280 [5.519 to 19.739]
  24 hours | 0.0000 [0.000 to 0.118] | 0.1050 [0.000 to 0.113] | 0.2620 [0.136 to 0.626] | 0.4790 [0.348 to 0.577] | 1.2020 [0.598 to 3.960] | 1.1015 [0.630 to 2.452] | 1.5040 [0.471 to 4.065]
  48 hours | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | 0.0000 [0.000 to 0.249] | 0.0000 [0.000 to 0.205] | 0.3440 [0.000 to 1.447] | 0.1895 [0.000 to 0.922] | 0.2565 [0.000 to 1.659]

47. Secondary Outcome: Part B: Plasma Concentrations of GSK3206944
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of GSK3206944. GSK3206944 is a metabolite of GSK3358699.
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

48. Secondary Outcome: Part C: Plasma Concentrations of GSK3206944
Description: as for outcome 46
Time Frame: as for outcome 27
Population: as for outcome 27
Measure: Median (Full Range); unit: Nanogram per milliliter
Arm/Group | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 RD | Part C: Cohort 7- GSK3358699 RD | Part C: Cohort 8- GSK3358699 RD
Number analyzed (Participants) | 14 | 0 | 0 | 0
Nanogram per milliliter
  Day 1:Pre-dose,n=14,0,0,0 | 0.0000 [0.000 to 0.000] |  |  |
  Day 1:15 minutes,n=14,0,0,0 | 0.0000 [0.000 to 0.459] |  |  |
  Day 1:30 minutes,n=14,0,0,0 | 3.1310 [0.116 to 12.947] |  |  |
  Day 1:1 hour,n=14,0,0,0 | 19.9335 [5.173 to 38.568] |  |  |
  Day 1:2 hours,n=14,0,0,0 | 22.2250 [11.285 to 56.829] |  |  |
  Day 1:4 hours,n=14,0,0,0 | 12.7730 [7.948 to 39.355] |  |  |
  Day 1:6 hours,n=14,0,0,0 | 7.2920 [4.588 to 18.565] |  |  |
  Day 1:8 hours,n=14,0,0,0 | 4.3750 [2.446 to 10.040] |  |  |
  Day 1:12 hours,n=14,0,0,0 | 2.2070 [0.883 to 4.176] |  |  |
  Day 1:24 hours,n=14,0,0,0 | 0.3805 [0.309 to 1.062] |  |  |
  Day 4: Pre-dose,n=14,0,0,0 | 0.5355 [0.000 to 0.890] |  |  |
  Day 8: Pre-dose,n=7,0,0,0: number analyzed (Participants) | 7 | 0 | 0 | 0
  Day 8: Pre-dose,n=7,0,0,0 | 0.6640 [0.200 to 1.233] |  |  |
  Day 12: Pre-dose,n=4,0,0,0: number analyzed (Participants) | 4 | 0 | 0 | 0
  Day 12: Pre-dose,n=4,0,0,0 | 0.4945 [0.382 to 1.217] |  |  |
  Day 14:Pre-dose,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:Pre-dose,n=2,0,0,0 | 0.5820 [0.549 to 0.615] |  |  |
  Day 14:15 minutes,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:15 minutes,n=2,0,0,0 | 0.7430 [0.582 to 0.904] |  |  |
  Day 14:30 minutes,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:30 minutes,n=2,0,0,0 | 6.4130 [4.906 to 7.920] |  |  |
  Day 14:1 hour,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:1 hour,n=2,0,0,0 | 15.3355 [14.722 to 15.949] |  |  |
  Day 14:2 hours,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:2 hours,n=2,0,0,0 | 15.0925 [14.474 to 15.711] |  |  |
  Day 14:4 hours,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:4 hours,n=2,0,0,0 | 10.4550 [9.880 to 11.030] |  |  |
  Day 14:6 hours,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:6 hours,n=2,0,0,0 | 6.8500 [5.834 to 7.866] |  |  |
  Day 14:8 hours,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:8 hours,n=2,0,0,0 | 6.0330 [3.779 to 8.287] |  |  |
  Day 14:12 hours,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:12 hours,n=2,0,0,0 | 2.2290 [1.424 to 3.034] |  |  |
  Day 14:24 hours,n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14:24 hours,n=2,0,0,0 | 0.5275 [0.445 to 0.610] |  |  |
  Day 14:48 hours,n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 14:48 hours,n=1,0,0,0 | 0.1110 [0.111 to 0.111] |  |  |

49. Secondary Outcome: Part A: AUC(0-t) of GSK3206944
Description: as for outcome 46
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population.
Measure: Median (Full Range); unit: Hours*nanogram per milliliter
Arm/Group | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 5 | 3 | 6 | 6 | 12 | 6 | 6
Hours*nanogram per milliliter | 15.16 [9.0 to 22.6] | 29.12 [25.0 to 31.6] | 106.55 [73.3 to 143.0] | 209.98 [172.2 to 376.7] | 381.16 [289.5 to 431.4] | 470.40 [403.1 to 706.8] | 630.63 [432.5 to 1030.1]

50. Secondary Outcome: Part B: AUC(0-t) of GSK3206944
Description: as for outcome 47
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

51. Secondary Outcome: Part C: AUC(0-t) of GSK3206944
Description: as for outcome 46
Time Frame: as for outcome 30
Population: as for outcome 27
Measure: Median (Full Range); unit: Hours*nanogram per milliliter
Arm/Group | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 RD | Part C: Cohort 7- GSK3358699 RD | Part C: Cohort 8- GSK3358699 RD
Number analyzed (Participants) | 14 | 0 | 0 | 0
Hours*nanogram per milliliter
  Day 1, n=14,0,0,0 | 115.17 [68.7 to 272.0] |  |  |
  Day 14, n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14, n=2,0,0,0 | 109.71 [94.7 to 124.7] |  |  |

52. Secondary Outcome: Part A: AUC(0-infinity) of GSK3206944
Description: as for outcome 46
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours*nanogram per milliliter
Arm/Group | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 2 | 2 | 6 | 4 | 8 | 4 | 6
Hours*nanogram per milliliter | 17.08 [16.4 to 17.8] | 29.05 [25.7 to 32.4] | 108.29 [74.7 to 144.3] | 189.02 [174.4 to 221.8] | 357.98 [291.8 to 419.1] | 492.92 [408.6 to 709.6] | 649.74 [443.5 to 1030.9]

53. Secondary Outcome: Part B: AUC(0-infinity) of GSK3206944
Description: as for outcome 47
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

54. Secondary Outcome: Part C: AUC(0-infinity) of GSK3206944
Description: as for outcome 46
Time Frame: as for outcome 30
Population: as for outcome 27
Measure: Median (Full Range); unit: Hours*nanogram per milliliter
Arm/Group | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 RD | Part C: Cohort 7- GSK3358699 RD | Part C: Cohort 8- GSK3358699 RD
Number analyzed (Participants) | 14 | 0 | 0 | 0
Hours*nanogram per milliliter
  Day 1, n=14,0,0,0 | 117.25 [71.2 to 274.6] |  |  |
  Day 14, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0

55. Secondary Outcome: Part A: AUC(0-24) of GSK3206944
Description: as for outcome 46
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours*nanogram per milliliter
Arm/Group | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 2 | 2 | 6 | 6 | 12 | 6 | 6
Hours*nanogram per milliliter | 16.44 [15.2 to 17.7] | 28.27 [25.0 to 31.6] | 106.55 [65.4 to 143.0] | 209.96 [172.2 to 368.7] | 374.49 [278.6 to 406.3] | 452.66 [377.9 to 692.4] | 586.70 [407.2 to 1019.2]

56. Secondary Outcome: Part B: AUC(0-24) of GSK3206944
Description: as for outcome 47
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

57. Secondary Outcome: Part C: AUC(0-24) of GSK3206944
Description: as for outcome 46
Time Frame: Days 1 and 14: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, and 24 hours post-dose
Population: as for outcome 27
Measure: Median (Full Range); unit: Hours*nanogram per milliliter
Arm/Group | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 RD | Part C: Cohort 7- GSK3358699 RD | Part C: Cohort 8- GSK3358699 RD
Number analyzed (Participants) | 14 | 0 | 0 | 0
Hours*nanogram per milliliter
  Day 1, n=14,0,0,0 | 115.31 [68.8 to 272.2] |  |  |
  Day 14, n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14, n=2,0,0,0 | 106.19 [94.7 to 117.7] |  |  |

58. Secondary Outcome: Part A: Cmax of GSK3206944
Description: as for outcome 46
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population.
Measure: Median (Full Range); unit: Nanogram per milliliter
Arm/Group | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 5 | 3 | 6 | 6 | 12 | 6 | 6
Nanogram per milliliter | 3.28 [2.1 to 4.9] | 6.03 [4.8 to 7.3] | 19.39 [7.6 to 30.5] | 50.13 [27.5 to 82.3] | 71.67 [44.3 to 105.1] | 102.09 [51.5 to 206.0] | 121.22 [88.3 to 231.7]

59. Secondary Outcome: Part B: Cmax of GSK3206944
Description: as for outcome 47
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

60. Secondary Outcome: Part C: Cmax of GSK3206944
Description: as for outcome 46
Time Frame: as for outcome 30
Population: as for outcome 27
Measure: Median (Full Range); unit: Nanogram per milliliter
Arm/Group | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 RD | Part C: Cohort 7- GSK3358699 RD | Part C: Cohort 8- GSK3358699 RD
Number analyzed (Participants) | 14 | 0 | 0 | 0
Nanogram per milliliter
  Day 1, n=14,0,0,0 | 23.02 [11.3 to 56.8] |  |  |
  Day 14, n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14, n=2,0,0,0 | 15.34 [14.7 to 15.9] |  |  |

61. Secondary Outcome: Part A: Tmax of GSK3206944
Description: as for outcome 46
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 5 | 3 | 6 | 6 | 12 | 6 | 6
Hours | 1.00 [1.0 to 2.0] | 2.00 [1.0 to 2.0] | 2.00 [1.0 to 2.0] | 2.01 [1.0 to 2.1] | 2.00 [2.0 to 4.0] | 2.00 [1.0 to 2.0] | 2.00 [1.0 to 2.0]

62. Secondary Outcome: Part B: Tmax of GSK3206944
Description: as for outcome 47
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

63. Secondary Outcome: Part C: Tmax of GSK3206944
Description: as for outcome 46
Time Frame: as for outcome 30
Population: as for outcome 27
Measure: Median (Full Range); unit: Hours
Arm/Group | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 RD | Part C: Cohort 7- GSK3358699 RD | Part C: Cohort 8- GSK3358699 RD
Number analyzed (Participants) | 14 | 0 | 0 | 0
Hours
  Day 1, n=14,0,0,0 | 2.00 [1.0 to 2.0] |  |  |
  Day 14, n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14, n=2,0,0,0 | 0.99 [0.98 to 1.0] |  |  |

64. Secondary Outcome: Part A: t1/2 of GSK3206944
Description: as for outcome 46
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 2 | 2 | 6 | 4 | 8 | 4 | 6
Hours | 4.97 [2.8 to 7.1] | 4.91 [4.8 to 5.0] | 4.10 [3.0 to 14.5] | 3.80 [3.5 to 4.3] | 7.81 [3.8 to 11.6] | 6.98 [4.1 to 8.8] | 6.76 [3.0 to 15.2]

65. Secondary Outcome: Part B: t1/2 of GSK3206944
Description: as for outcome 47
Time Frame: Day 1: Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

66. Secondary Outcome: Part C: t1/2 of GSK3206944
Description: as for outcome 46
Time Frame: as for outcome 30
Population: as for outcome 27
Measure: Median (Full Range); unit: Hours
Arm/Group | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 RD | Part C: Cohort 7- GSK3358699 RD | Part C: Cohort 8- GSK3358699 RD
Number analyzed (Participants) | 14 | 0 | 0 | 0
Hours
  Day 1, n=14,0,0,0 | 5.02 [3.3 to 5.6] |  |  |
  Day 14, n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 14, n=2,0,0,0 | 6.15 [5.5 to 6.8] |  |  |

67. Secondary Outcome: Part A: Monocyte Intracellular Concentration of GSK3206944
Description: Blood samples were collected into sodium heparin tubes for the isolation of monocytes and for measurement of GSK3206944 concentrations in monocytes. GSK3206944 is a metabolite of GSK3358699.
Time Frame: Day 1: 1, 4, 8, 24 and 48 hours post-dose in each treatment period
Population: PK Population.
Measure: Median (Full Range); unit: Nanogram per milliliter
Arm/Group | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 5 | 3 | 6 | 6 | 12 | 6 | 6
Nanogram per milliliter
  Day 1: 1 hour | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | 0.177 [0.00 to 0.60] | 0.673 [0.00 to 1.08] | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | 1.243 [0.63 to 2.13] | 1.410 [0.94 to 1.94]
  Day 1: 4 hours | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | 0.105 [0.00 to 0.26] | 0.149 [0.00 to 0.84] | 0.277 [0.00 to 0.38] | 0.297 [0.00 to 0.45]
  Day 1: 8 hours | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification.
  Day 1: 24 hours | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification.
  Day 1: 48 hours | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification.

68. Secondary Outcome: Part B: Monocyte Intracellular Concentration of GSK3206944
Description: Blood samples were planned to be collected into sodium heparin tubes for the isolation of monocytes and for measurement of GSK3206944 concentrations in monocytes. GSK3206944 is a metabolite of GSK3358699.
Time Frame: Day 1: 1, 4, 8, 24 and 48 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

69. Secondary Outcome: Part C: Monocyte Intracellular Concentration of GSK3206944
Description: as for outcome 67
Time Frame: Days 1 and 13: 1, 4 and 8 hour; Days 4, 8 and 12: Pre-dose; Day 14: 1, 4, 8, 24 and 48 hours post-dose
Population: as for outcome 27
Measure: Median (Full Range); unit: Nanogram per milliliter
Arm/Group | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 RD | Part C: Cohort 7- GSK3358699 RD | Part C: Cohort 8- GSK3358699 RD
Number analyzed (Participants) | 14 | 0 | 0 | 0
Nanogram per milliliter
  Day 1: 1 hour,n=14,0,0,0 | 0.313 [0.00 to 0.56] |  |  |
  Day 1: 4 hours,n=14,0,0,0 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. |  |  |
  Day 1: 8 hours,n=14,0,0,0 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. |  |  |
  Day 4: Pre-dose,n=14,0,0,0 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. |  |  |
  Day 8: Pre-dose,n=14,0,0,0 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. |  |  |
  Day 12: Pre-dose,n=14,0,0,0 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. |  |  |
  Day 13: 1 hour,n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 13: 1 hour,n=1,0,0,0 | 0.317 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual monocyte intracellular concentration for this single participant. |  |  |
  Day 13: 4 hours,n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 13: 4 hours,n=1,0,0,0 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. |  |  |
  Day 13: 8 hours,n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 13: 8 hours,n=1,0,0,0 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. |  |  |
  Day 14: 1 hour,n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 14: 1 hour,n=1,0,0,0 | 0.256 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual monocyte intracellular concentration for this single participant. |  |  |
  Day 14: 4 hours,n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 14: 4 hours,n=1,0,0,0 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. |  |  |
  Day 14: 8 hours,n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 14: 8 hours,n=1,0,0,0 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. |  |  |
  Day 14: 24 hours,n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 14: 24 hours,n=1,0,0,0 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. |  |  |
  Day 14: 48 hours,n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 14: 48 hours,n=1,0,0,0 | NA [NA to NA] — Data could not be calculated as it was below the limit of quantification. |  |  |

70. Secondary Outcome: Part A: Absolute Values of Monocyte Chemotactic Protein (MCP)-1, Interleukin (IL)6, Tumor Necrosis Factor (TNF) Alpha in Blood After Ex-vivo Lipopolysaccharide (LPS) Activation
Description: Whole blood samples of 1 milliliter (mL) were collected in TruCulture tubes, containing LPS and incubated for 24 hours, post which the inflammatory mediators (MCP-1, IL-6 and TNF alpha) were analyzed.
Time Frame: Day 1: 1, 4, 8, 12, 24 and 48 hours
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles). Data was not collected for GSK3358699 25 mg SD arm.
Measure: Median (Full Range); unit: Picogram per milliliter
Arm/Group | Part A: Placebo SD | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD
Number analyzed (Participants) | 17 | 5 | 3 | 6 | 6 | 0 | 6 | 6
Picogram per milliliter
  Day 1: IL6, 1 hour, n=17,5,3,6,6,0,6,6 | 10352.87 [6166.6 to 19166.3] | 15208.12 [7257.3 to 24940.9] | 20385.25 [13064.2 to 22017.3] | 12820.72 [9166.6 to 33445.0] | 15596.95 [3426.4 to 28751.1] |  | 10057.64 [5014.4 to 17359.8] | 5728.17 [4267.2 to 18422.7]
  Day 1: IL6, 4 hours, n=17,5,3,6,6,0,6,6 | 13092.01 [4833.9 to 19117.2] | 13851.61 [9601.7 to 23110.3] | 19431.61 [16293.4 to 24387.6] | 15636.75 [8048.6 to 34008.3] | 12900.07 [6507.3 to 25108.1] |  | 12074.28 [4669.2 to 21515.6] | 7544.02 [5345.9 to 26788.0]
  Day 1: IL6, 8 hours, n=17,5,3,6,6,0,6,6 | 12560.83 [7112.0 to 33941.2] | 13629.60 [10440.1 to 27946.6] | 28805.81 [24272.2 to 31362.4] | 16564.79 [11058.8 to 26785.4] | 17019.48 [12120.4 to 21106.7] |  | 16486.96 [7413.4 to 21952.6] | 8688.63 [6758.8 to 20765.0]
  Day 1: IL6, 12 hour, n=17,5,3,6,6,0,6,6 | 15125.82 [2587.2 to 26028.6] | 13890.39 [11271.0 to 21279.4] | 28948.13 [24063.6 to 33176.4] | 18712.82 [6493.7 to 26803.1] | 15622.25 [10623.8 to 24243.3] |  | 12305.88 [8132.7 to 19539.9] | 6754.46 [3909.8 to 13207.0]
  Day 1: IL6, 24 hours, n=17,5,3,6,6,0,6,6 | 12876.74 [5221.8 to 19587.8] | 16961.79 [10045.9 to 23511.8] | 23634.22 [17018.1 to 32159.5] | 14387.39 [9362.7 to 32140.8] | 12593.53 [8519.9 to 32945.4] |  | 12894.02 [5914.3 to 17523.1] | 8705.59 [6150.6 to 23530.0]
  Day 1: IL6, 48 hours, n=17,5,3,6,6,0,6,6 | 13204.84 [6897.8 to 24379.3] | 16209.14 [8492.7 to 25387.3] | 27160.99 [17882.7 to 45604.5] | 14786.71 [10321.9 to 33336.3] | 13685.44 [7729.6 to 20697.6] |  | 14374.44 [8079.6 to 19835.0] | 8359.81 [6088.1 to 19757.4]
  Day 1: MCP-1, 1 hour, n=17,5,2,6,6,0,6,6: number analyzed (Participants) | 17 | 5 | 2 | 6 | 6 | 0 | 6 | 6
  Day 1: MCP-1, 1 hour, n=17,5,2,6,6,0,6,6 | 2107.38 [692.3 to 4748.1] | 2997.62 [775.1 to 5062.0] | 2539.15 [1560.9 to 3517.4] | 1273.19 [872.5 to 2047.4] | 1278.42 [640.5 to 2640.6] |  | 1604.85 [863.0 to 3331.4] | 1047.32 [716.5 to 1933.0]
  Day 1: MCP-1, 4 hours, n=17,5,3,6,6,0,6,6 | 1748.71 [878.2 to 3917.7] | 2638.95 [1272.7 to 2942.2] | 3774.02 [2841.1 to 4578.7] | 1410.01 [617.5 to 1973.0] | 1648.51 [559.9 to 4038.0] |  | 2604.00 [918.1 to 3465.2] | 1643.37 [1067.0 to 3385.4]
  Day 1: MCP-1, 8 hours, n=17,5,3,6,6,0,6,6 | 1300.34 [713.0 to 3074.7] | 2911.87 [1297.8 to 4926.4] | 3145.66 [2964.7 to 3966.5] | 1606.85 [993.1 to 2784.3] | 1533.33 [634.0 to 3454.9] |  | 2312.12 [899.7 to 3203.8] | 1863.25 [1295.9 to 3392.0]
  Day 1: MCP-1, 12 hour, n=17,5,3,6,6,0,6,6 | 1791.07 [808.9 to 4505.9] | 2738.20 [2017.5 to 4140.2] | 3048.56 [3045.4 to 4036.5] | 2003.41 [832.7 to 4276.2] | 1297.53 [903.3 to 5483.9] |  | 2062.41 [1546.5 to 3811.4] | 2270.49 [882.1 to 7042.9]
  Day 1: MCP-1, 24 hours, n=17,5,3,6,6,0,6,6 | 1662.28 [673.9 to 3360.2] | 2349.62 [912.1 to 3608.3] | 2216.41 [1124.8 to 5178.2] | 1691.59 [661.1 to 2299.7] | 1062.86 [369.0 to 5821.6] |  | 2275.17 [845.9 to 2731.8] | 1988.64 [1360.9 to 3313.2]
  Day 1: MCP-1, 48 hours, n=17,5,3,6,6,0,6,6 | 1398.36 [526.2 to 4408.1] | 2306.83 [577.0 to 4174.3] | 1621.46 [1505.3 to 3215.7] | 1729.87 [958.5 to 2877.5] | 1200.15 [514.4 to 3554.8] |  | 1595.51 [1082.1 to 2315.4] | 1828.23 [894.9 to 2434.1]
  Day 1: TNF alpha, 1 hour, n=17,5,3,6,6,0,6,6 | 2525.78 [1073.6 to 4950.0] | 2281.20 [2214.6 to 5283.6] | 4340.00 [2395.2 to 6512.0] | 3455.53 [2172.3 to 12708.3] | 3916.76 [567.9 to 5873.5] |  | 1971.77 [992.6 to 3554.9] | 1552.10 [640.6 to 5120.6]
  Day 1: TNF alpha, 4 hours, n=17,5,3,6,6,0,6,6 | 3189.81 [1264.1 to 5492.9] | 3452.27 [3139.9 to 8159.2] | 3381.52 [3014.8 to 8775.2] | 4493.55 [1481.7 to 16761.7] | 2672.58 [1527.3 to 7834.4] |  | 3618.72 [698.0 to 5482.5] | 1876.55 [1429.5 to 10939.6]
  Day 1: TNF alpha, 8 hours, n=17,5,3,6,6,0,6,6 | 3673.78 [1891.2 to 8758.2] | 3630.47 [2520.6 to 8206.4] | 9631.19 [8462.1 to 9881.2] | 4612.79 [2513.7 to 10996.7] | 4908.42 [3867.7 to 7647.1] |  | 5233.22 [1875.8 to 6062.3] | 2934.21 [2142.3 to 8128.1]
  Day 1: TNF alpha, 12 hour, n=17,5,3,6,6,0,6,6 | 4206.18 [717.0 to 9209.7] | 3680.34 [3268.1 to 6257.6] | 8736.93 [7805.2 to 10949.6] | 5139.53 [1199.2 to 10251.4] | 3079.37 [2178.8 to 7014.1] |  | 2846.57 [1964.6 to 7505.2] | 1729.42 [1203.4 to 2845.9]
  Day 1: TNF alpha, 24 hours, n=17,5,3,5,6,0,6,6: number analyzed (Participants) | 17 | 5 | 3 | 5 | 6 | 0 | 6 | 6
  Day 1: TNF alpha, 24 hours, n=17,5,3,5,6,0,6,6 | 3164.79 [845.9 to 6087.5] | 4528.14 [3348.7 to 7098.2] | 4694.58 [3321.5 to 13261.4] | 5576.01 [1699.4 to 12223.1] | 3543.62 [2185.0 to 9815.1] |  | 3649.08 [1319.2 to 4891.2] | 2741.96 [1683.3 to 8477.3]
  Day 1: TNF alpha, 48 hours, n=17,5,3,6,6,0,6,6 | 3445.95 [2189.6 to 7880.2] | 4077.77 [2120.7 to 6772.6] | 10364.95 [3942.4 to 14023.2] | 4186.10 [2069.1 to 12454.5] | 3963.40 [1613.3 to 5663.8] |  | 3788.04 [2727.4 to 5746.1] | 2404.11 [1734.5 to 6985.8]

71. Secondary Outcome: Part B: Absolute Values of MCP-1, IL6, TNF Alpha in Blood After Ex-vivo LPS Activation
Description: Whole blood samples were planned to be collected in TruCulture tubes, containing LPS and incubated for 24 hours, post which the inflammatory mediators (MCP-1, IL6 and TNF alpha) were planned to be analyzed.
Time Frame: Day 1: 1, 4, 8, 12, 24 and 48 hours
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed
Number analyzed (Participants) | 0 | 0

72. Secondary Outcome: Part C: Absolute Values of MCP-1, IL6, TNF Alpha in Blood After Ex-vivo LPS Activation
Description: Whole blood samples of 1 mL were collected in TruCulture tubes, containing LPS and incubated for 24 hours, post which the inflammatory mediators (MCP-1, IL-6 and TNF alpha) were analyzed.
Time Frame: Day 1: 1, 4 and 8 hours; Days 2, 4, 8 and 12: Pre-dose; Day 13: Pre-dose, 1, 4 and 8 hours; Day 14: Pre-dose, Pre-LPS challenge, 1, 4, 8, 24 and 48 hours
Population: Safety Population. Data was not collected for Cohorts 6 to 8 as no participants were enrolled. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Median (Full Range); unit: Picogram per milliliter
Groups:
- Part C: Cohort 4 and 5- Placebo RD: Participants received once daily RD of placebo on Days 1 to 14. In Cohort 4, on Day 14, participants were administered an IV in vivo LPS challenge at a dose of 0.75 ng/kg or an IV infusion of GM-CSF, in vivo at a dose of 60 mcg/m^2. The administration of LPS or GM CSF was followed by blister induction on forearm (0.2% cantharidin).
- Part C: Cohort 4 and 5- GSK3358699 10 mg RD: Participants received once daily repeat dose of GSK3358699 10 mg on Days 1 to 14. In Cohort 4, on Day 14, participants were administered an IV in vivo LPS challenge at a dose of 0.75 ng/kg or an IV infusion of GM-CSF, in vivo at a dose of 60 mcg/m^2. The administration of LPS or GM CSF was followed by blister induction on forearm (0.2% cantharidin).
- Part C: Cohort 8- GSK3358699 or Placebo RD: Participants in Part C Cohort 8 were planned to receive once daily repeat dose of GSK3358699 or placebo on Days 1 to 14. On Day 14, participants were planned to receive an IV in vivo LPS challenge at a dose of 0.75 ng/kg or an IV infusion of GM-CSF, in vivo as 60 mcg/m^2. The administration of LPS or GM CSF was planned to be followed by blister induction on forearm (0.2% cantharidin).
Arm/Group | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
Number analyzed (Participants) | 11 | 14 | 0 | 0 | 0
Picogram per milliliter
  IL6:Day 1,1 hour,n=11,13,0,0,0: number analyzed (Participants) | 11 | 13 | 0 | 0 | 0
  IL6:Day 1,1 hour,n=11,13,0,0,0 | 9488.65 [331.7 to 16540.5] | 9629.75 [3513.3 to 14975.4] |  |  |
  IL6:Day 1,4 hours,n=11,14,0,0,0 | 9121.35 [3866.4 to 18996.3] | 10686.75 [3976.0 to 17276.8] |  |  |
  IL6:Day 1,8 hours,n=11,14,0,0,0 | 13079.21 [5597.2 to 20424.0] | 15475.58 [1340.7 to 35210.3] |  |  |
  IL6:Day 2,Pre-dose,n=11,14,0,0,0 | 9323.67 [4126.4 to 19011.4] | 12396.71 [5456.9 to 19819.0] |  |  |
  IL6:Day 4,Pre-dose,n=11,14,0,0,0 | 11002.47 [2713.4 to 19232.1] | 12558.78 [4188.7 to 20344.2] |  |  |
  IL6:Day 8,Pre-dose,n=6,7,0,0,0: number analyzed (Participants) | 6 | 7 | 0 | 0 | 0
  IL6:Day 8,Pre-dose,n=6,7,0,0,0 | 11305.84 [8590.8 to 31436.0] | 10766.02 [4511.8 to 13171.8] |  |  |
  IL6:Day 12,Pre-dose,n=5,4,0,0,0: number analyzed (Participants) | 5 | 4 | 0 | 0 | 0
  IL6:Day 12,Pre-dose,n=5,4,0,0,0 | 9329.36 [7777.5 to 16845.5] | 10539.82 [7378.2 to 12671.6] |  |  |
  IL6:Day 13,Pre-dose,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  IL6:Day 13,Pre-dose,n=1,1,0,0,0 | 9966.64 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. | 12743.26 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. |  |  |
  IL6:Day 13,1 hour,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  IL6:Day 13,1 hour,n=1,1,0,0,0 | 11718.40 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. | 12508.94 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. |  |  |
  IL6:Day 13,4 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  IL6:Day 13,4 hours,n=1,1,0,0,0 | 7099.42 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. | 11616.53 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. |  |  |
  IL6:Day 13,8 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  IL6:Day 13,8 hours,n=1,1,0,0,0 | 10722.24 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. | 16723.58 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. |  |  |
  IL6:Day 14,Pre-dose,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  IL6:Day 14,Pre-dose,n=1,1,0,0,0 | 8918.96 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. | 14654.83 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. |  |  |
  IL6:Day 14,Pre LPS challenge,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  IL6:Day 14,Pre LPS challenge,n=1,1,0,0,0 | 8696.65 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. | 11340.79 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. |  |  |
  IL6:Day 14,1 hour,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  IL6:Day 14,1 hour,n=1,1,0,0,0 | 10082.23 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. | 13244.20 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. |  |  |
  IL6:Day 14,4 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  IL6:Day 14,4 hours,n=1,1,0,0,0 | 9122.21 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. | 11543.08 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. |  |  |
  IL6:Day 14,8 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  IL6:Day 14,8 hours,n=1,1,0,0,0 | 10986.16 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. | 12544.55 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. |  |  |
  IL6:Day 14,24 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  IL6:Day 14,24 hours,n=1,1,0,0,0 | 9176.89 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. | 9114.15 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. |  |  |
  IL6:Day 14,48 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  IL6:Day 14,48 hours,n=1,1,0,0,0 | 8257.88 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. | 10304.01 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual IL6 for this single participant. |  |  |
  MCP-1:Day 1,1 hour,n=11,14,0,0,0 | 1739.49 [114.6 to 4212.9] | 2216.06 [1080.4 to 4084.7] |  |  |
  MCP-1:Day 1,4 hours,n=11,14,0,0,0 | 1825.09 [813.5 to 3719.8] | 2405.11 [996.0 to 5337.9] |  |  |
  MCP-1:Day 1,8 hours,n=11,14,0,0,0 | 2002.44 [656.7 to 4982.8] | 2044.64 [148.3 to 2887.4] |  |  |
  MCP-1:Day 2,Pre-dose,n=11,14,0,0,0 | 1939.09 [511.6 to 4614.3] | 1928.51 [818.2 to 4090.7] |  |  |
  MCP-1:Day 4,Pre-dose,n=11,14,0,0,0 | 1677.88 [537.9 to 3500.9] | 1939.65 [747.5 to 3428.4] |  |  |
  MCP-1:Day 8,Pre-dose,n=6,7,0,0,0: number analyzed (Participants) | 6 | 7 | 0 | 0 | 0
  MCP-1:Day 8,Pre-dose,n=6,7,0,0,0 | 1638.33 [1129.3 to 6091.9] | 1719.26 [1336.5 to 3634.5] |  |  |
  MCP-1:Day 12,Pre-dose,n=5,4,0,0,0: number analyzed (Participants) | 5 | 4 | 0 | 0 | 0
  MCP-1:Day 12,Pre-dose,n=5,4,0,0,0 | 1799.12 [1262.3 to 4483.2] | 2176.12 [497.9 to 2954.5] |  |  |
  MCP-1:Day 13,Pre-dose,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  MCP-1:Day 13,Pre-dose,n=1,1,0,0,0 | 1839.00 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. | 513.36 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. |  |  |
  MCP-1:Day 13,1 hour,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  MCP-1:Day 13,1 hour,n=1,1,0,0,0 | 2113.92 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. | 294.72 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. |  |  |
  MCP-1:Day 13,4 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  MCP-1:Day 13,4 hours,n=1,1,0,0,0 | 1872.12 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. | 890.77 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. |  |  |
  MCP-1:Day 13,8 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  MCP-1:Day 13,8 hours,n=1,1,0,0,0 | 1997.87 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. | 1412.52 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. |  |  |
  MCP-1:Day 14,Pre-dose,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  MCP-1:Day 14,Pre-dose,n=1,1,0,0,0 | 2007.09 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. | 4935.03 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. |  |  |
  MCP-1:Day 14,Pre LPS challenge,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  MCP-1:Day 14,Pre LPS challenge,n=1,1,0,0,0 | 1876.05 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. | 1981.15 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. |  |  |
  MCP-1:Day 14,1 hour,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  MCP-1:Day 14,1 hour,n=1,1,0,0,0 | 3503.11 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. | 3623.79 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. |  |  |
  MCP-1:Day 14,4 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  MCP-1:Day 14,4 hours,n=1,1,0,0,0 | 2066.72 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. | 3293.92 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. |  |  |
  MCP-1:Day 14,8 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  MCP-1:Day 14,8 hours,n=1,1,0,0,0 | 2593.90 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. | 3150.84 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. |  |  |
  MCP-1:Day 14,24 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  MCP-1:Day 14,24 hours,n=1,1,0,0,0 | 2082.28 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. | 3372.94 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. |  |  |
  MCP-1:Day 14,48 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  MCP-1:Day 14,48 hours,n=1,1,0,0,0 | 1879.53 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. | 2715.94 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual MCP-1 for this single participant. |  |  |
  TNF alpha:Day 1,1 hour,n=11,13,0,0,0: number analyzed (Participants) | 11 | 13 | 0 | 0 | 0
  TNF alpha:Day 1,1 hour,n=11,13,0,0,0 | 1994.72 [135.2 to 3287.3] | 2078.66 [962.5 to 4069.3] |  |  |
  TNF alpha:Day 1,4 hours,n=11,14,0,0,0 | 1843.08 [596.4 to 4580.6] | 2297.36 [1173.8 to 4818.4] |  |  |
  TNF alpha:Day 1,8 hours,n=11,14,0,0,0 | 3692.36 [1094.9 to 6402.9] | 3854.86 [289.5 to 13254.5] |  |  |
  TNF alpha:Day 2,Pre-dose,n=11,14,0,0,0 | 2711.07 [849.2 to 4558.3] | 3028.33 [1506.6 to 5961.8] |  |  |
  TNF alpha:Day 4,Pre-dose,n=11,14,0,0,0 | 2987.24 [456.6 to 5033.0] | 3045.05 [1202.4 to 5443.8] |  |  |
  TNF alpha:Day 8,Pre-dose,n=6,7,0,0,0: number analyzed (Participants) | 6 | 7 | 0 | 0 | 0
  TNF alpha:Day 8,Pre-dose,n=6,7,0,0,0 | 2932.72 [2616.4 to 7598.9] | 2849.52 [784.2 to 3366.7] |  |  |
  TNF alpha:Day 12,Pre-dose,n=5,4,0,0,0: number analyzed (Participants) | 5 | 4 | 0 | 0 | 0
  TNF alpha:Day 12,Pre-dose,n=5,4,0,0,0 | 2482.03 [1958.2 to 3588.4] | 2407.60 [1143.7 to 2971.6] |  |  |
  TNF alpha:Day 13,Pre-dose,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  TNF alpha:Day 13,Pre-dose,n=1,1,0,0,0 | 2311.66 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. | 2995.36 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. |  |  |
  TNF alpha:Day 13,1 hour,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  TNF alpha:Day 13,1 hour,n=1,1,0,0,0 | 3495.21 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. | 2648.27 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. |  |  |
  TNF alpha:Day 13,4 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  TNF alpha:Day 13,4 hours,n=1,1,0,0,0 | 1573.18 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. | 2815.39 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. |  |  |
  TNF alpha:Day 13,8 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  TNF alpha:Day 13,8 hours,n=1,1,0,0,0 | 2486.89 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. | 4472.25 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. |  |  |
  TNF alpha:Day 14,Pre-dose,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  TNF alpha:Day 14,Pre-dose,n=1,1,0,0,0 | 2304.40 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. | 3327.69 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. |  |  |
  TNF alpha:Day 14,Pre LPS challenge,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  TNF alpha:Day 14,Pre LPS challenge,n=1,1,0,0,0 | 2092.07 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. | 2081.54 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. |  |  |
  TNF alpha:Day 14,1 hour,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  TNF alpha:Day 14,1 hour,n=1,1,0,0,0 | 2103.62 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. | 3133.32 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. |  |  |
  TNF alpha:Day 14,4 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  TNF alpha:Day 14,4 hours,n=1,1,0,0,0 | 1771.69 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. | 2457.35 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. |  |  |
  TNF alpha:Day 14,8 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  TNF alpha:Day 14,8 hours,n=1,1,0,0,0 | 2560.84 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. | 3481.91 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. |  |  |
  TNF alpha:Day 14,24 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  TNF alpha:Day 14,24 hours,n=1,1,0,0,0 | 1482.94 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. | 2187.40 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. |  |  |
  TNF alpha:Day 14,48 hours,n=1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  TNF alpha:Day 14,48 hours,n=1,1,0,0,0 | 1909.65 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. | 2597.32 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual TNF alpha for this single participant. |  |  |

ADVERSE EVENTS:
Time Frame: Up to Day 193 in Part A and up to Day 49 in Part C (Cohorts 4 and 5)
Description: Safety Population.All-cause mortality,non-SAEs and SAEs were not collected in Part B and Part C(Cohorts 6 to 8) as no participants were enrolled.Data is presented for Part A and Part C(Cohorts4 and 5) only as data was not collected in Part B and Part C(Cohorts6 to 8) due to study termination and Part B and Part C(Cohorts 6 to 8) were not initiated.
Arm/Group | Part A: Placebo SD | Part A: GSK3358699 1 mg SD | Part A: GSK3358699 3 mg SD | Part A: GSK3358699 10 mg SD | Part A: GSK3358699 20 mg SD | Part A: GSK3358699 25 mg SD | Part A: GSK3358699 30 mg SD | Part A: GSK3358699 40 mg SD | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed | Part C: Cohort 4 and 5- Placebo RD | Part C: Cohort 4 and 5- GSK3358699 10 mg RD | Part C: Cohort 6- GSK3358699 or Placebo RD | Part C: Cohort 7- GSK3358699 or Placebo RD | Part C: Cohort 8- GSK3358699 or Placebo RD
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/5 | 0/3 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/0 | 0/0 | 0/11 | 0/14 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/5 | 0/3 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/0 | 0/0 | 0/11 | 1/14 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 4/23 | 2/5 | 3/3 | 2/6 | 3/6 | 8/12 | 4/6 | 3/6 | 0/0 | 0/0 | 7/11 | 7/14 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo SD (N=23) | Part A: GSK3358699 1 mg SD (N=5) | Part A: GSK3358699 3 mg SD (N=3) | Part A: GSK3358699 10 mg SD (N=6) | Part A: GSK3358699 20 mg SD (N=6) | Part A: GSK3358699 25 mg SD (N=12) | Part A: GSK3358699 30 mg SD (N=6) | Part A: GSK3358699 40 mg SD (N=6) | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted (N=0) | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed (N=0) | Part C: Cohort 4 and 5- Placebo RD (N=11) | Part C: Cohort 4 and 5- GSK3358699 10 mg RD (N=14) | Part C: Cohort 6- GSK3358699 or Placebo RD (N=0) | Part C: Cohort 7- GSK3358699 or Placebo RD (N=0) | Part C: Cohort 8- GSK3358699 or Placebo RD (N=0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo SD (N=23) | Part A: GSK3358699 1 mg SD (N=5) | Part A: GSK3358699 3 mg SD (N=3) | Part A: GSK3358699 10 mg SD (N=6) | Part A: GSK3358699 20 mg SD (N=6) | Part A: GSK3358699 25 mg SD (N=12) | Part A: GSK3358699 30 mg SD (N=6) | Part A: GSK3358699 40 mg SD (N=6) | Part B: Cohort 3- GSK3358699 Fed + GSK3358699 Fasted (N=0) | Part B: Cohort 3- GSK3358699 Fasted + GSK3358699 Fed (N=0) | Part C: Cohort 4 and 5- Placebo RD (N=11) | Part C: Cohort 4 and 5- GSK3358699 10 mg RD (N=14) | Part C: Cohort 6- GSK3358699 or Placebo RD (N=0) | Part C: Cohort 7- GSK3358699 or Placebo RD (N=0) | Part C: Cohort 8- GSK3358699 or Placebo RD (N=0)
Headache (Nervous system disorders) | 2 (2) | 1 (3) | 1 (1) | 1 (3) | 2 (2) | 4 (4) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal atrophy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT03426995/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT03426995/SAP_001.pdf